CLINICAL TRIAL: NCT02315066
Title: A PHASE 1, OPEN-LABEL, DOSE ESCALATION STUDY OF PF-04518600 AS A SINGLE AGENT AND IN COMBINATION WITH PF-05082566 IN PATIENTS WITH SELECTED LOCALLY ADVANCED OR METASTATIC CANCERS
Brief Title: Study Of OX40 Agonist PF-04518600 Alone And In Combination With 4-1BB Agonist PF-05082566
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B0601002; 2014-004107-75 (EudraCT Number); B0601002 (Other: Alias Study Number); OX40 (Other: Alias Study Number)
Record Dates: First submitted 2014-12-04; First posted 2014-12-11 (Estimated); Results first posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-02

CONDITIONS: Neoplasms
Keywords: Immunotherapy; PF-04518600; PF-05082566; solid tumors; tumors; neoplasm metastasis; Phase 1; hepatocellular carcinoma; HCC; liver cancer; ocular melanoma; melanoma; clear cell renal cell carcinoma; RCC; kidney cancer; head and neck squamous cell carcinoma; HNSCC; head and neck cancer; cervical cancer; cancer of the cervix; gastric cancer; stomach cancer; non small cell lung cancer; NSCLC; lung cancer; urothelial bladder carcinoma; bladder cancer; OX40; 4-1BB
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Carcinoma, Hepatocellular; Liver Neoplasms; Uveal Melanoma; Melanoma; Carcinoma, Renal Cell; Kidney Neoplasms; Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Uterine Cervical Neoplasms; Stomach Neoplasms; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Urinary Bladder Neoplasms | interventions — utomilumab

STUDY DESIGN:
Masking Description: Open-label
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-04518600 (Experimental): OX40 agonist
  Interventions: Drug: PF-04518600
- PF-04518600 plus PF-05082566 (Experimental): OX40 (CD134) agonist plus 4-1BB (CD137) agonist
  Interventions: Drug: PF-04518600 plus PF-05082566

INTERVENTIONS:
Drug: PF-04518600 — Part A1 - PF-04518600 will be administered intravenously every 14 days in cohorts of 2 or more patients starting at a dose of 0.01 mg/kg. Increases in dose will continue until MTD is determined
  Arms: PF-04518600
Drug: PF-04518600 — Part A2 - patients with hepatocellular carcinoma will be randomized to receive treatment with PF-04518600 at various doses administered intravenously
  Arms: PF-04518600
Drug: PF-04518600 plus PF-05082566 — Part B1 -In cohorts of 2 or more patients, PF-04518600 will be administered intravenously every 2 weeks starting at a dose of 0.1 mg/kg and PF-05082566 will be administered intravenously 4 weeks starting at a dose of 20 mg. Increases in dose will continue until MTD is determined.
  Arms: PF-04518600 plus PF-05082566
Drug: PF-04518600 plus PF-05082566 — Part B2 - patients with select tumor types (ocular melanoma, cutaneous/acral melanoma or non-small cell lung cancer) will be treated at dose levels based on the OBD selected in Part 1.
  Arms: PF-04518600 plus PF-05082566

SUMMARY:
To assess the safety and tolerability at increasing dose levels of PF-04518600 alone or in combination wtih PF-05082566 in patients with select advanced or metastatic carcinoma in order to determine the maximum tolerated dose and select the recommended Phase 2 dose.

ELIGIBILITY:
Inclusion Criteria:

* Part A1 only: Patients with histological or cytological diagnosis of HNSCC, HCC, melanoma, or clear cell RCC who progressed on or are intolerant to standard therapy, for which no standard therapy is available or who decline standard therapy.
* Part A2 only: Patients with histological or cytological diagnosis of advanced/metastatic HCC who are treatment naïve and have declined standard of care, or have had at least 1 prior line of systemic therapy. Prior anti PD L1/PD 1 therapy is allowed.
* Part B1 only: Patients with histological or cytological diagnosis of NSCLC, HNSCC, melanoma, urothelial bladder carcinoma (including renal pelvis, ureters, urinary bladder, and urethra), gastric or squamous cell carcinoma of the uterine cervix who progressed on or are intolerant to standard therapy, for which no standard therapy is available, or who decline standard therapy.
* Part B2

Arm 1 only:

1. Ocular melanoma patients with advanced/metastatic disease, or
2. Cutaneous/acral melanoma patients with advanced/metastatic disease who have received checkpoint inhibitor (anti PD L1, anti PD 1, or anti CTLA4) based treatment on which disease progressed. [Note: Checkpoint inhibitor may have been part of a combination therapy, as long as the combination did not contain OX40 or 4 1BB agonist.] Any questions on prior treatment may be discussed with the Sponsor.

Arm 2 only:

* Histological or cytological diagnosis of NSCLC with advanced/metastatic disease. Patients must have previously received prior anti PD L1 or anti PD 1 mAb on which disease progressed. [Note: Previous anti PD L1 or anti PD 1 mAb may have been part of a combination therapy, eg, in combination with chemotherapy, as long as the combination did not contain OX40 or 4 1BB agonist.]
* Performance Status of 0 or 1 - Adequate bone marrow, kidney and liver function

Exclusion Criteria:

* Brain metastases requiring steroids
* Major surgery, Radiation therapy within 4 weeks of starting study treatment (except: palliative radiotherapy to a limited field is allowed after consultation with sponsor's medical monitor at any time during study participation, including during screening), or systemic anti-cancer therapy within 4 weeks of study treatment start (6 weeks for mitomycin C or nitrosoureas)
* Active and clinically significant bacterial, fungal, or viral infection
* History of active autoimmune disorders
* History of immune-mediated adverse events requiring immunosuppressive therapy or were grade 3 or higher related to prior immune-modulatory therapy
* Prior treatment with an OX40 agonist and 4-1BB agonist (for Part B1/B2)
* Prior anthracycline treatment and at risk of cardiac failure (New York Heart Association Class 2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2015-04-23 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (30):
- United States (24):
  - The Angeles Clinic And Research Institute, A Cedars-Sinai Affiliate, Los Angeles, California
  - Keck Hospital of USC, Los Angeles, California
  - LAC+USC Medical Center, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Ronald Regan Medical Center, Los Angeles, California
  - UCLA Hematology & Oncology Clinic, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Medical Imaging Center of Southern California, Inc., Santa Monica, California
  - Santa Monica UCLA Hematology & Oncology Clinic, Santa Monica, California
  - UConn Health, Pharmacy, Farmington, Connecticut
  - UConn Health, Neag Comprehensive Cancer Center, Farmington, Connecticut
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Massachusetts General Hospital (MGH), Boston, Massachusetts
  - Brigham & Women's Hospital (BWH), Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (BIDMC), Boston, Massachusetts
  - Dana-Farber Cancer Institute (DFCI), Boston, Massachusetts
  - Massachusetts General/Chelsea HealthCare Center, Chelsea, Massachusetts
  - Mass General/North Shore Center for Outpatient Care, Danvers, Massachusetts
  - Mass General West, Waltham, Massachusetts
  - Columbia University Medical Center - Herbert Irving Pavilion, New York, New York
  - Methodist Hospital-Pathology, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- France (2):
  - Groupe hospitalier Pitie Salpetriere, Paris
  - Institut Gustave Roussy, Villejuif
- National Cancer Center Hospital East, Kashiwa, Chiba, Japan
- Netherlands (3):
  - The Netherlands Cancer Institute, Amsterdam
  - Slotervaart Hospital/Antoni van Leeuwenhoek, Amsterdam
  - Erasmus MC, Rotterdam

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Hamid O, Chiappori AA, Thompson JA, Doi T, Hu-Lieskovan S, Eskens FALM, Ros W, Diab A, Spano JP, Rizvi NA, Wasser JS, Angevin E, Ott PA, Forgie A, Yang W, Guo C, Chou J, El-Khoueiry AB. First-in-human study of an OX40 (ivuxolimab) and 4-1BB (utomilumab) agonistic antibody combination in patients with advanced solid tumors. J Immunother Cancer. 2022 Oct;10(10):e005471. doi: 10.1136/jitc-2022-005471. PMID 36302562
- [Derived] Diab A, Hamid O, Thompson JA, Ros W, Eskens FALM, Doi T, Hu-Lieskovan S, Klempner SJ, Ganguly B, Fleener C, Wang X, Joh T, Liao K, Salek-Ardakani S, Taylor CT, Chou J, El-Khoueiry AB. A Phase I, Open-Label, Dose-Escalation Study of the OX40 Agonist Ivuxolimab in Patients with Locally Advanced or Metastatic Cancers. Clin Cancer Res. 2022 Jan 1;28(1):71-83. doi: 10.1158/1078-0432.CCR-21-0845. Epub 2021 Oct 6. PMID 34615725
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0601002&StudyName=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part A (PF-04518600 monotherapy) included Part A1 and Part A2 Part B(PF-04518600 plus utomilumab [PF-05082566] combination therapy) included Part B1 and Part B2
Pre-assignment Details: A total of 174 participants were enrolled in this study, and 174 of them received study treatment. For Part A, 87 participants were enrolled and treated with PF-04518600 at several dose levels. For Part B, 87 participants were enrolled and treated with PF-04518600+utomilumab at several dose levels.
Groups:
- Part A1: PF-04518600 0.01mg/kg: Participants received PF-04518600 0.01mg/kg IV over about 60 minutes on Day 1 of each cycle of 2 weeks up to a maximum of 14 weeks.
- Part A1: PF-04518600 0.1mg/kg: Participants received PF-04518600 0.1mg/kg IV over about 60 minutes on Day 1 of each cycle of 2 weeks up to a maximum of 14 weeks.
- Part A1: PF-04518600 0.3mg/kg: Participants received PF-04518600 0.3mg/kg IV over about 60 minutes on Day 1 of each cycle of 2 weeks up to a maximum of 14 weeks.
- Part A1: PF-04518600 1.5mg/kg: Participants received PF-04518600 1.5mg/kg IV over about 60 minutes on Day 1 of each cycle of 2 weeks up to a maximum of 14 weeks.
- Part A1: PF-04518600 3.0mg/kg: Participants received PF-04518600 3.0mg/kg IV over about 60 minutes on Day 1 of each cycle of 2 weeks up to a maximum of 14 weeks.
- Part A1: PF-04518600 10mg/kg: Participants received PF-04518600 10mg/kg IV over about 60 minutes on Day 1 of each cycle of 2 weeks up to a maximum of 14 weeks.
- Part A2: PF-04518600 30mg: Participants received PF-04518600 30mg IV over about 60 minutes on Day 1 of each cycle of 2 weeks up to a maximum of 14 weeks.
- Part A2: PF-04518600 250mg: Participants received PF-04518600 250mg IV over about 60 minutes on Day 1 of each cycle of 2 weeks up to a maximum of 14 weeks.
- Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg: Participants received PF-05082566 20mg IV over about 60 minutes on Day 1 of every 28 days and PF-04518600 0.1mg/kg IV over about 60 minutes on Day 1 of each cycle of 2 weeks. On cycles whereby both PF-04518600 and PF-05082566 were to be administered on the same day, PF-04518600 were administered after, but no sooner than 30 minutes after completion of the PF-05082566 infusion in absence of infusion reaction and after post PF-05082566 and pre PF-04518600 pharmacokinetic blood draws.
- Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg: Participants received PF-05082566 20mg IV over about 60 minutes on Day 1 of every 28 days and PF-04518600 0.3mg/kg IV over about 60 minutes on Day 1 of each cycle of 2 weeks. On cycles whereby both PF-04518600 and PF-05082566 were to be administered on the same day, PF-04518600 were administered after, but no sooner than 30 minutes after completion of the PF-05082566 infusion in absence of infusion reaction and after post PF-05082566 and pre PF-04518600 pharmacokinetic blood draws.
- Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg: Participants received PF-05082566 100mg IV over about 60 minutes on Day 1 of every 28 days and PF-04518600 0.3mg/kg IV over about 60 minutes on Day 1 of each cycle of 2 weeks. On cycles whereby both PF-04518600 and PF-05082566 were to be administered on the same day, PF-04518600 were administered after, but no sooner than 30 minutes after completion of the PF-05082566 infusion in absence of infusion reaction and after post PF-05082566 and pre PF-04518600 pharmacokinetic blood draws.
- Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg: Participants received PF-05082566 100mg IV over about 60 minutes on Day 1 of every 28 days and PF-04518600 1.0mg/kg IV over about 60 minutes on Day 1 of each cycle of 2 weeks. On cycles whereby both PF-04518600 and PF-05082566 were to be administered on the same day, PF-04518600 were administered after, but no sooner than 30 minutes after completion of the PF-05082566 infusion in absence of infusion reaction and after post PF-05082566 and pre PF-04518600 pharmacokinetic blood draws.
- Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg: Participants received PF-05082566 100mg IV over about 60 minutes on Day 1 of every 28 days and PF-04518600 3.0mg/kg IV over about 60 minutes on Day 1 of each cycle of 2 weeks. On cycles whereby both PF-04518600 and PF-05082566 were to be administered on the same day, PF-04518600 were administered after, but no sooner than 30 minutes after completion of the PF-05082566 infusion in absence of infusion reaction and after post PF-05082566 and pre PF-04518600 pharmacokinetic blood draws.
- Part B2: PF-04518600 30mg + PF-05082566 20mg: Participants received PF-05082566 20mg IV over about 60 minutes on Day 1 of every 28 days and PF-04518600 30mg IV over about 60 minutes on Day 1 of each cycle of 2 weeks. On cycles whereby both PF-04518600 and PF-05082566 were to be administered on the same day, PF-04518600 were administered after, but no sooner than 30 minutes after completion of the PF-05082566 infusion in absence of infusion reaction and after post PF-05082566 and pre PF-04518600 pharmacokinetic blood draws.
Period: Overall Study
Arm/Group | Part A1: PF-04518600 0.01mg/kg | Part A1: PF-04518600 0.1mg/kg | Part A1: PF-04518600 0.3mg/kg | Part A1: PF-04518600 1.5mg/kg | Part A1: PF-04518600 3.0mg/kg | Part A1: PF-04518600 10mg/kg | Part A2: PF-04518600 30mg | Part A2: PF-04518600 250mg | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg | Part B2: PF-04518600 30mg + PF-05082566 20mg
Started | 2 | 10 | 11 | 12 | 13 | 4 | 16 | 19 | 11 | 12 | 12 | 11 | 11 | 30
Completed | 0 | 0 | 2 | 1 | 2 | 1 | 3 | 5 | 0 | 1 | 0 | 0 | 1 | 0
Not Completed | 2 | 10 | 9 | 11 | 11 | 3 | 13 | 14 | 11 | 11 | 12 | 11 | 10 | 30
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 2 | 0 | 4
Not completed — Death | 2 | 7 | 6 | 11 | 10 | 3 | 9 | 9 | 10 | 8 | 10 | 7 | 8 | 21
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Subject refused further follow-up | 0 | 2 | 2 | 0 | 0 | 0 | 2 | 3 | 0 | 1 | 1 | 2 | 2 | 4
Not completed — Study ongoing at date of cut-off | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all enrolled patients who received at least one full or partial IV infusion of study drug PF-04518600.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A1: PF-04518600 0.01mg/kg | Part A1: PF-04518600 0.1mg/kg | Part A1: PF-04518600 0.3mg/kg | Part A1: PF-04518600 1.5mg/kg | Part A1: PF-04518600 3.0mg/kg | Part A1: PF-04518600 10mg/kg | Part A2: PF-04518600 30mg | Part A2: PF-04518600 250mg | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg | Part B2: PF-04518600 30mg + PF-05082566 20mg | Total
Number analyzed (Participants) | 2 | 10 | 11 | 12 | 13 | 4 | 16 | 19 | 11 | 12 | 12 | 11 | 11 | 30 | 174
Age, Customized [Number; unit: participants]
  Less than 18 years old | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18 to 44 years old (18-44) | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 3 | 11
  45 to 64 years old (45-64) | 2 | 7 | 6 | 2 | 7 | 1 | 8 | 9 | 7 | 7 | 8 | 4 | 3 | 14 | 85
  65 years old and more than 65 years old (>＝65) | 0 | 2 | 3 | 10 | 6 | 2 | 8 | 9 | 2 | 5 | 3 | 7 | 8 | 13 | 78
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3 | 1 | 2 | 0 | 0 | 3 | 4 | 4 | 7 | 3 | 9 | 10 | 49
  Male | 1 | 8 | 8 | 11 | 11 | 4 | 16 | 16 | 7 | 8 | 5 | 8 | 2 | 20 | 125
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 0 | 1 | 0 | 1 | 0 | 2 | 2 | 4 | 1 | 0 | 0 | 2 | 16
  Not Hispanic or Latino | 2 | 7 | 11 | 11 | 13 | 3 | 8 | 14 | 9 | 8 | 11 | 11 | 11 | 24 | 143
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 3 | 0 | 0 | 0 | 0 | 0 | 4 | 15
Race/Ethnicity, Customized [Number; unit: participants]
  WHITE | 1 | 10 | 9 | 9 | 8 | 4 | 6 | 8 | 10 | 6 | 10 | 8 | 8 | 20 | 117
  BLACK | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 6
  ASIAN | 0 | 0 | 1 | 3 | 4 | 0 | 2 | 5 | 1 | 2 | 2 | 3 | 3 | 4 | 30
  OTHER | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 4 | 0 | 0 | 0 | 3 | 10
  UNSPECIFIED | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 11
Body mass index [Mean (Standard Deviation); unit: kilograms per meter squared (kg/m^2)] | 27.5 (6.7) | 26.6 (3.6) | 26.4 (4.9) | 28.9 (5.7) | 25.9 (4.5) | 22.8 (1.9) | 26.2 (3.7) | 25.5 (6.0) | 25.3 (5.2) | 26.7 (7.6) | 25.5 (7.4) | 25.0 (5.2) | 23.5 (5.9) | 25.2 (5.3) | 25.2 (5.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) in Part A1
Description: DLT was defined as any of the following adverse events occurring in the first two cycle of treatment (28 days), unless there was a clear alternative explanation: hematologic: grade 4 neutropenia lasting >7 days, febrile neutropenia; grade ≥3 neutropenic infection; grade ≥3 thrombocytopenia with clinically significant bleeding or requiring medical intervention; grade 4 thrombocytopenia; grade 4 anemia; grade ≥3 anemia related to hemolysis or autoimmune disease. non hematologic: grade ≥3 toxicities that were considered clinically significant, including cytokine release syndrome, infusion reactions and allergic reactions, except those that had not been maximally treated or could be easily treated. The severity of adverse events was graded as per common terminology criteria for adverse events(CTCAE) version 4.03, and there were no DLTs reported.
Time Frame: The first 2 cycles of treatment (Day 1 up to Day 28)
Population: The population for this outcome measure included all enrolled participants who received at least two cycles of study medication and who did not have major treatment deviations during first two cycles.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A1: PF-04518600 0.01mg/kg | Part A1: PF-04518600 0.1mg/kg | Part A1: PF-04518600 0.3mg/kg | Part A1: PF-04518600 1.5mg/kg | Part A1: PF-04518600 3.0mg/kg | Part A1: PF-04518600 10mg/kg
Number analyzed (Participants) | 2 | 10 | 11 | 12 | 13 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With All-Causality Treatment Emergent Adverse Events(TEAEs) and Serious Adverse Event(SAEs), Treatment-Related TEAEs and SAEs in Part A
Description: Adverse event (AE) was graded by the investigator according to CTCAE version 4.03 and coded using the Medical Dictionary for Regulatory Activities (MedDRA): Grade 3 (Severe) events=unacceptable or intolerable events. Grade 4 (Life-threatening) events caused participant to be in imminent danger of death. Grade 5 (Death) events=death related to an AE. Treatment-emergent events=between first dose of study drug and up to 35 days after last dose that were absent before treatment or that worsened relative to pretreatment state. TEAEs were defined as those with initial onset or increasing in severity after the first dose of study medication. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: AEs: The informed consent date up to the last dosing date + 28 days or all drug-related toxicities resolved date. SAEs: The informed consent date through first dosing date + 98 days or up to the last dosing date + 60 days, and any post-reporting period.
Population: Analysis population included all enrolled participants who received at least one full or partial IV infusion of study drug PF-04518600.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A1: PF-04518600 0.01mg/kg | Part A1: PF-04518600 0.1mg/kg | Part A1: PF-04518600 0.3mg/kg | Part A1: PF-04518600 1.5mg/kg | Part A1: PF-04518600 3.0mg/kg | Part A1: PF-04518600 10mg/kg | Part A2: PF-04518600 30mg | Part A2: PF-04518600 250mg
Number analyzed (Participants) | 2 | 10 | 11 | 12 | 13 | 4 | 16 | 19
Participants
  Number of Participants with all-causality TEAEs | 2 | 10 | 11 | 12 | 13 | 4 | 16 | 19
  Number of Participants with treatment-related TEAEs | 2 | 7 | 7 | 7 | 7 | 1 | 11 | 12
  Number of Participants with treatment-related SAEs | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
  Number of Participants with all-causality SAEs | 0 | 4 | 1 | 3 | 6 | 2 | 7 | 6

3. Primary Outcome: Number of Participants With Laboratory Test Abnormalities in Part A
Description: Following parameters were analyzed for laboratory examination: hematology (hemoglobin, hematocrit, platelet count, white blood cell count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes, partial thromboplastin time (PTT), Prothrombin (PT), PT international ratio); liver function (aspartate aminotransferase(AST), alanine aminotransferase(ALT), total bilirubin, gamma-glutamyl transpeptidase(GT), alkaline phosphatase, albumin, total protein); renal function (blood urea nitrogen, creatinine, uric acid); electrolytes (sodium, potassium, chloride, calcium , phosphate, magnesium); clinical chemistry (glucose, creatine kinase, thyroxine (T4), thyroid stimulating hormone(TSH)), Amylase, Lipase), urinalysis (dipstick [protein, blood], microscopy [urine red blood cell (RBC), white blood cell (WBC), Epithelial Cells], miscellaneous [urine casts and bacteria]).
Time Frame: The first dosing date to the earlier date between the last dosing date + 35 days and the first new anti-cancer therapy date (if applicable)
Population: Analysis Population included all enrolled participants who received at least 1 full or partial IV infusion of study drug PF-04518600.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A1: PF-04518600 0.01mg/kg | Part A1: PF-04518600 0.1mg/kg | Part A1: PF-04518600 0.3mg/kg | Part A1: PF-04518600 1.5mg/kg | Part A1: PF-04518600 3.0mg/kg | Part A1: PF-04518600 10mg/kg | Part A2: PF-04518600 30mg | Part A2: PF-04518600 250mg
Number analyzed (Participants) | 2 | 10 | 11 | 12 | 12 | 4 | 16 | 19
Participants
  Hemoglobin (g/dL) < 0.8 x lower limit of normal (LLN) | 0 | 2 | 4 | 6 | 4 | 2 | 10 | 4
  Hematocrit (%) < 0.8 x LLN: number analyzed (Participants) | 2 | 9 | 9 | 11 | 10 | 4 | 16 | 19
  Hematocrit (%) < 0.8 x LLN | 0 | 1 | 2 | 4 | 5 | 3 | 8 | 5
  Platelets (10**3/mm**3) < 0.5 x LLN | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Platelets (10**3/mm**3) > 1.75 x upper limit of normal (ULN) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White Blood Cell Count (10**3/mm**3) < 0.6 x LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  White Blood Cell Count (10**3/mm**3) > 1.5 x ULN | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0
  Lymphocytes (Absolute(Abs)) (10**3/mm**3) < 0.8 x LLN: number analyzed (Participants) | 2 | 8 | 9 | 12 | 11 | 4 | 10 | 17
  Lymphocytes (Absolute(Abs)) (10**3/mm**3) < 0.8 x LLN | 1 | 2 | 2 | 5 | 4 | 4 | 6 | 8
  Lymphocytes (Abs) (10**3/mm**3) > 1.2 x ULN: number analyzed (Participants) | 2 | 8 | 9 | 12 | 11 | 4 | 10 | 17
  Lymphocytes (Abs) (10**3/mm**3) > 1.2 x ULN | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1
  Lymphocytes (%) < 0.8 x LLN: number analyzed (Participants) | 2 | 9 | 9 | 11 | 10 | 4 | 16 | 19
  Lymphocytes (%) < 0.8 x LLN | 2 | 7 | 5 | 7 | 9 | 4 | 9 | 10
  Lymphocytes (%) > 1.2 x ULN: number analyzed (Participants) | 2 | 9 | 9 | 11 | 10 | 4 | 16 | 19
  Lymphocytes (%) > 1.2 x ULN | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
  Total Neutrophils (Abs) (10**3/mm**3) < 0.8 x LLN: number analyzed (Participants) | 2 | 10 | 11 | 12 | 12 | 4 | 15 | 18
  Total Neutrophils (Abs) (10**3/mm**3) < 0.8 x LLN | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3
  Total Neutrophils (Abs) (10**3/mm**3) > 1.2 x LLN: number analyzed (Participants) | 2 | 10 | 11 | 12 | 12 | 4 | 15 | 18
  Total Neutrophils (Abs) (10**3/mm**3) > 1.2 x LLN | 0 | 1 | 1 | 2 | 6 | 3 | 1 | 5
  Neutrophils (%) <0.8x LLN: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 19
  Neutrophils (%) <0.8x LLN |  |  |  |  |  |  | 0 | 0
  Neutrophils (%) >1.2x ULN: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 19
  Neutrophils (%) >1.2x ULN |  |  |  |  |  |  | 1 | 3
  PTT (sec) > 1.1 x ULN: number analyzed (Participants) | 2 | 9 | 10 | 11 | 10 | 4 | 16 | 19
  PTT (sec) > 1.1 x ULN | 2 | 2 | 4 | 4 | 3 | 1 | 3 | 4
  Basophils (Abs) (10**3/mm**3) > 1.2 x ULN: number analyzed (Participants) | 2 | 8 | 9 | 11 | 11 | 4 | 9 | 17
  Basophils (Abs) (10**3/mm**3) > 1.2 x ULN | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 0
  Basophils (%) > 1.2 x ULN: number analyzed (Participants) | 2 | 9 | 9 | 11 | 10 | 4 | 16 | 19
  Basophils (%) > 1.2 x ULN | 0 | 2 | 3 | 1 | 2 | 1 | 2 | 4
  Eosinophils (Abs) (10**3/mm**3) > 1.2 x ULN: number analyzed (Participants) | 2 | 8 | 9 | 11 | 11 | 4 | 9 | 17
  Eosinophils (Abs) (10**3/mm**3) > 1.2 x ULN | 1 | 0 | 3 | 1 | 3 | 0 | 2 | 2
  Eosinophils (%) > 1.2 x ULN: number analyzed (Participants) | 2 | 9 | 9 | 11 | 10 | 4 | 16 | 19
  Eosinophils (%) > 1.2 x ULN | 1 | 3 | 7 | 4 | 3 | 1 | 4 | 6
  Monocytes (Abs) (10**3/mm**3) > 1.2 x ULN: number analyzed (Participants) | 2 | 8 | 9 | 11 | 11 | 4 | 9 | 17
  Monocytes (Abs) (10**3/mm**3) > 1.2 x ULN | 0 | 2 | 3 | 4 | 2 | 3 | 0 | 3
  Monocytes (%) > 1.2 x ULN: number analyzed (Participants) | 2 | 9 | 9 | 11 | 10 | 4 | 16 | 19
  Monocytes (%) > 1.2 x ULN | 1 | 4 | 3 | 10 | 8 | 1 | 5 | 12
  Prothrombin (PT) (sec) > 1.1 x ULN | 0 | 0 | 2 | 5 | 2 | 2 | 4 | 6
  PT International Ratio (INR) > 1.1 x ULN | 0 | 0 | 2 | 5 | 1 | 0 | 5 | 6
  Total Bilirubin (mg/dL) > 1.5 x ULN | 1 | 3 | 0 | 1 | 2 | 0 | 5 | 5
  Direct Bilirubin (mg/dL) > 1.5 x ULN: number analyzed (Participants) | 1 | 0 | 1 | 1 | 1 | 1 | 3 | 5
  Direct Bilirubin (mg/dL) > 1.5 x ULN | 1 |  | 0 | 1 | 1 | 0 | 3 | 4
  Indirect Bilirubin (mg/dL) > 1.5 x ULN: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 4
  Indirect Bilirubin (mg/dL) > 1.5 x ULN |  |  |  | 0 |  | 0 | 0 | 1
  Aspartate Aminotransferase (AST) (IU/L) > 3.0 x ULN | 1 | 4 | 0 | 3 | 3 | 0 | 6 | 9
  Alanine Aminotransferase (ALT) (IU/L) > 3.0 x ULN | 0 | 2 | 0 | 1 | 2 | 0 | 4 | 5
  Gamma GT (IU/L) > 3.0 x ULN: number analyzed (Participants) | 0 | 3 | 3 | 6 | 8 | 4 | 16 | 19
  Gamma GT (IU/L) > 3.0 x ULN |  | 1 | 0 | 4 | 4 | 0 | 10 | 10
  Alkaline Phosphatase (IU/L) > 3.0 x ULN | 0 | 3 | 0 | 4 | 3 | 0 | 5 | 7
  Albumin (g/dL) < 0.8 x LLN | 0 | 0 | 1 | 4 | 2 | 2 | 1 | 4
  Albumin (g/dL) > 1.2 x ULN | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Blood Urea Nitrogen (BUN) (mg/dL) > 1.3 x ULN | 1 | 2 | 2 | 3 | 4 | 0 | 2 | 1
  Creatinine (mg/dL) > 1.3 x ULN | 0 | 1 | 2 | 1 | 3 | 0 | 1 | 2
  Uric Acid (mg/dL) > 1.2 x ULN | 0 | 3 | 2 | 2 | 3 | 1 | 2 | 4
  Sodium (milliequivalent (mEq/L) < 0.95 x LLN | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 2
  Sodium (mEq/L) > 1.05 x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium (mEq/L) < 0.9 x LLN | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Potassium (mEq/L) > 1.1 x ULN | 0 | 1 | 0 | 1 | 3 | 0 | 1 | 0
  Chloride (mEq/L) < 0.9 x LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chloride (mEq/L) > 1.1 x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium (mg/dL) < 0.9 x LLN | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 0
  Calcium (mg/dL) > 1.1 x ULN | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
  Magnesium (mg/dL) < 0.9 x LLN | 1 | 1 | 0 | 3 | 2 | 1 | 0 | 1
  Magnesium (mg/dL) > 1.1 x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Phosphate (mg/dL) < 0.8 x LLN | 0 | 0 | 1 | 0 | 1 | 2 | 3 | 3
  Phosphate (mg/dL) > 1.2 x ULN | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  T4 (free) (ng/dL) < 0.8 x LLN: number analyzed (Participants) | 0 | 1 | 1 | 4 | 3 | 3 | 9 | 14
  T4 (free) (ng/dL) < 0.8 x LLN |  | 0 | 0 | 0 | 0 | 0 | 0 | 0
  T4 (free) (ng/dL) > 1.2 x ULN: number analyzed (Participants) | 0 | 1 | 1 | 4 | 3 | 3 | 9 | 14
  T4 (free) (ng/dL) > 1.2 x ULN |  | 0 | 0 | 0 | 1 | 0 | 0 | 2
  TSH (UIU/mL) < 0.8 x LLN: number analyzed (Participants) | 0 | 1 | 2 | 4 | 6 | 4 | 15 | 19
  TSH (UIU/mL) < 0.8 x LLN |  | 0 | 0 | 0 | 0 | 0 | 1 | 1
  TSH (UIU/mL) > 1.2 x ULN: number analyzed (Participants) | 0 | 1 | 2 | 4 | 6 | 4 | 15 | 19
  TSH (UIU/mL) > 1.2 x ULN |  | 0 | 0 | 1 | 2 | 2 | 3 | 6
  Glucose (mg/dL) < 0.6 x LLN | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose (mg/dL) > 1.5 x ULN | 0 | 6 | 2 | 5 | 4 | 1 | 9 | 5
  Creatine Kinase (CK) (U/L) > 2.0 x ULN: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 4
  Creatine Kinase (CK) (U/L) > 2.0 x ULN |  |  | 0 | 0 |  |  | 0 | 0
  Amylase (U/L) > 1.5 x ULN | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 5
  Lipase (U/L) > 1.5 x ULN | 1 | 1 | 1 | 1 | 2 | 0 | 4 | 3
  Urine Protein (Qual) >= 1 | 1 | 5 | 4 | 4 | 1 | 1 | 5 | 5
  Urine Blood/ hemoglobin(Hgb) (Qual) >= 1 | 0 | 1 | 2 | 3 | 3 | 2 | 1 | 2
  Urine RBC (/high power field (HPF)) >= 20: number analyzed (Participants) | 1 | 10 | 11 | 12 | 12 | 4 | 16 | 19
  Urine RBC (/high power field (HPF)) >= 20 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 2
  Urine WBC (/HPF) >= 20: number analyzed (Participants) | 1 | 10 | 11 | 12 | 12 | 4 | 16 | 19
  Urine WBC (/HPF) >= 20 | 0 | 0 | 0 | 3 | 2 | 2 | 0 | 0
  Urine Epithelial Cells (/HPF) >= 6: number analyzed (Participants) | 1 | 8 | 8 | 10 | 11 | 3 | 5 | 13
  Urine Epithelial Cells (/HPF) >= 6 | 0 | 3 | 3 | 1 | 3 | 2 | 1 | 3
  Urine Casts (/low power field(LPF) > 1: number analyzed (Participants) | 1 | 4 | 7 | 4 | 5 | 1 | 6 | 4
  Urine Casts (/low power field(LPF) > 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Urine Granular Casts (/LPF) > 1: number analyzed (Participants) | 1 | 5 | 7 | 4 | 5 | 1 | 1 | 1
  Urine Granular Casts (/LPF) > 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
  Urine Hyaline Casts (/LPF) >1: number analyzed (Participants) | 1 | 6 | 8 | 7 | 8 | 2 | 2 | 6
  Urine Hyaline Casts (/LPF) >1 | 1 | 4 | 2 | 5 | 5 | 0 | 1 | 4
  Urine Bacteria (/HPF) > 20: number analyzed (Participants) | 1 | 9 | 9 | 11 | 11 | 2 | 7 | 16
  Urine Bacteria (/HPF) > 20 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With DLTs in Part B1
Description: as for outcome 1
Time Frame: The First 2 Cycles of Treatment (Day 1 up to Day 28)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 11
Participants | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With All-causality TEAEs and SAEs, and Treatment-Related TEAEs and SAEs in Part B
Description: as for outcome 2
Time Frame: AEs: The informed consent date up to the last dosing date + 60 days or all drug-related toxicities resolved date. SAEs: The informed consent date through first dosing date + 98 days or up to the last dosing date + 60 days, and any post-reporting period.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg | Part B2: PF-04518600 30mg + PF-05082566 20mg
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 11 | 30
Participants
  Number of Participants with all-causality TEAEs | 11 | 12 | 12 | 11 | 11 | 30
  Number of Participants with treatment-related TEAEs | 4 | 6 | 7 | 5 | 7 | 22
  Number of Participants with treatment-related SAEs | 0 | 0 | 0 | 1 | 0 | 0
  Number of Participants with all-causality SAEs | 5 | 2 | 3 | 5 | 5 | 10

6. Primary Outcome: Number of Participants With Laboratory Test Abnormalities in Part B
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg | Part B2: PF-04518600 30mg + PF-05082566 20mg
Number analyzed (Participants) | 10 | 12 | 12 | 11 | 11 | 30
Participants
  Hemoglobin (g/dL) < 0.8 x lower limit of normal (LLN) | 4 | 3 | 4 | 7 | 6 | 9
  Hematocrit (%) < 0.8 x LLN: number analyzed (Participants) | 9 | 10 | 10 | 10 | 11 | 29
  Hematocrit (%) < 0.8 x LLN | 4 | 2 | 3 | 6 | 4 | 4
  Platelets (10**3/mm**3) < 0.5 x LLN | 0 | 1 | 0 | 0 | 0 | 0
  Platelets (10**3/mm**3) > 1.75 x upper limit of normal (ULN) | 0 | 0 | 1 | 3 | 0 | 1
  White Blood Cell Count (10**3/mm**3) < 0.6 x LLN | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Count (10**3/mm**3) > 1.5 x ULN | 0 | 1 | 4 | 2 | 3 | 6
  Lymphocytes (Abs) (10**3/mm**3) < 0.8 x LLN: number analyzed (Participants) | 8 | 11 | 12 | 10 | 11 | 28
  Lymphocytes (Abs) (10**3/mm**3) < 0.8 x LLN | 5 | 5 | 8 | 6 | 6 | 10
  Lymphocytes (Abs) (10**3/mm**3) > 1.2 x ULN: number analyzed (Participants) | 8 | 11 | 12 | 10 | 11 | 28
  Lymphocytes (Abs) (10**3/mm**3) > 1.2 x ULN | 1 | 0 | 0 | 1 | 1 | 1
  Lymphocytes (%) < 0.8 x LLN: number analyzed (Participants) | 9 | 10 | 10 | 10 | 11 | 29
  Lymphocytes (%) < 0.8 x LLN | 8 | 8 | 9 | 9 | 9 | 20
  Lymphocytes (%) > 1.2 x ULN: number analyzed (Participants) | 9 | 10 | 10 | 10 | 11 | 29
  Lymphocytes (%) > 1.2 x ULN | 1 | 0 | 0 | 1 | 1 | 0
  Total Neutrophils (Abs) (10**3/mm**3) < 0.8 x LLN | 0 | 0 | 1 | 0 | 0 | 0
  Total Neutrophils (Abs) (10**3/mm**3) > 1.2 x LLN | 3 | 5 | 5 | 7 | 5 | 15
  Neutrophils (%) <0.8x LLN: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 29
  Neutrophils (%) <0.8x LLN |  |  |  |  |  | 2
  Neutrophils (%) >1.2x ULN: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 29
  Neutrophils (%) >1.2x ULN |  |  |  |  |  | 6
  Basophils (Abs) (10**3/mm**3) > 1.2 x ULN: number analyzed (Participants) | 8 | 11 | 12 | 10 | 11 | 28
  Basophils (Abs) (10**3/mm**3) > 1.2 x ULN | 0 | 0 | 0 | 0 | 0 | 5
  Basophils (%) > 1.2 x ULN: number analyzed (Participants) | 9 | 10 | 10 | 10 | 11 | 29
  Basophils (%) > 1.2 x ULN | 0 | 0 | 1 | 0 | 0 | 3
  Eosinophils (Abs) (10**3/mm**3) > 1.2 x ULN: number analyzed (Participants) | 8 | 11 | 12 | 10 | 11 | 28
  Eosinophils (Abs) (10**3/mm**3) > 1.2 x ULN | 1 | 3 | 6 | 4 | 3 | 12
  Eosinophils (%) > 1.2 x ULN: number analyzed (Participants) | 9 | 10 | 10 | 10 | 11 | 29
  Eosinophils (%) > 1.2 x ULN | 1 | 3 | 6 | 3 | 4 | 14
  Monocytes (Abs) (10**3/mm**3) > 1.2 x ULN: number analyzed (Participants) | 8 | 11 | 12 | 10 | 11 | 28
  Monocytes (Abs) (10**3/mm**3) > 1.2 x ULN | 1 | 4 | 5 | 6 | 5 | 9
  Monocytes (%) > 1.2 x ULN: number analyzed (Participants) | 9 | 10 | 10 | 10 | 11 | 29
  Monocytes (%) > 1.2 x ULN | 3 | 3 | 3 | 6 | 3 | 9
  PTT (sec) > 1.1 x ULN: number analyzed (Participants) | 9 | 11 | 10 | 11 | 11 | 29
  PTT (sec) > 1.1 x ULN | 3 | 1 | 3 | 4 | 2 | 7
  Prothrombin (PT) (sec) > 1.1 x ULN: number analyzed (Participants) | 10 | 12 | 12 | 10 | 11 | 30
  Prothrombin (PT) (sec) > 1.1 x ULN | 1 | 3 | 2 | 3 | 3 | 11
  PT International Ratio (INR) > 1.1 x ULN: number analyzed (Participants) | 10 | 11 | 12 | 9 | 11 | 30
  PT International Ratio (INR) > 1.1 x ULN | 2 | 1 | 0 | 0 | 1 | 3
  Total Bilirubin (mg/dL) > 1.5 x ULN | 0 | 0 | 1 | 0 | 1 | 0
  Direct Bilirubin (mg/dL) > 1.5 x ULN: number analyzed (Participants) | 0 | 1 | 3 | 1 | 1 | 2
  Direct Bilirubin (mg/dL) > 1.5 x ULN |  | 0 | 1 | 0 | 0 | 0
  Indirect Bilirubin (mg/dL) > 1.5 x ULN: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 1
  Indirect Bilirubin (mg/dL) > 1.5 x ULN |  |  | 0 |  | 0 | 0
  Aspartate Aminotransferase (AST) (IU/L) > 3.0 x ULN | 0 | 0 | 1 | 0 | 2 | 1
  Alanine Aminotransferase (ALT) (IU/L) > 3.0 x ULN | 0 | 0 | 1 | 0 | 0 | 3
  Gamma GT (IU/L) > 3.0 x ULN | 1 | 0 | 2 | 2 | 2 | 5
  Alkaline Phosphatase (IU/L) > 3.0 x ULN | 1 | 0 | 1 | 1 | 1 | 1
  Albumin (g/dL) < 0.8 x LLN | 1 | 0 | 2 | 3 | 3 | 3
  Albumin (g/dL) > 1.2 x ULN | 0 | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen (BUN) (mg/dL) > 1.3 x ULN | 1 | 2 | 2 | 1 | 1 | 5
  Creatinine (mg/dL) > 1.3 x ULN | 1 | 1 | 3 | 0 | 1 | 2
  Uric Acid (mg/dL) > 1.2 x ULN | 1 | 1 | 0 | 0 | 2 | 1
  Sodium (mEq/L) < 0.95 x LLN | 0 | 1 | 0 | 1 | 3 | 2
  Sodium (mEq/L) > 1.05 x ULN | 0 | 0 | 0 | 0 | 0 | 0
  Potassium (mEq/L) < 0.9 x LLN | 0 | 0 | 2 | 0 | 1 | 1
  Potassium (mEq/L) > 1.1 x ULN | 0 | 0 | 1 | 0 | 1 | 5
  Chloride (mEq/L) < 0.9 x LLN | 0 | 1 | 1 | 0 | 1 | 1
  Chloride (mEq/L) > 1.1 x ULN | 0 | 0 | 0 | 0 | 0 | 0
  Calcium (mg/dL) < 0.9 x LLN | 1 | 0 | 1 | 1 | 1 | 1
  Calcium (mg/dL) > 1.1 x ULN | 0 | 0 | 0 | 2 | 1 | 0
  Magnesium (mg/dL) < 0.9 x LLN | 1 | 1 | 4 | 2 | 1 | 3
  Magnesium (mg/dL) > 1.1 x ULN | 0 | 1 | 0 | 0 | 0 | 0
  Phosphate (mg/dL) < 0.8 x LLN | 0 | 0 | 2 | 0 | 1 | 2
  Phosphate (mg/dL) > 1.2 x ULN | 0 | 0 | 0 | 0 | 0 | 0
  T4 (free) (ng/dL) < 0.8 x LLN: number analyzed (Participants) | 4 | 7 | 7 | 8 | 6 | 13
  T4 (free) (ng/dL) < 0.8 x LLN | 0 | 0 | 0 | 0 | 0 | 0
  T4 (free) (ng/dL) > 1.2 x ULN: number analyzed (Participants) | 4 | 7 | 7 | 8 | 6 | 13
  T4 (free) (ng/dL) > 1.2 x ULN | 0 | 0 | 0 | 0 | 1 | 1
  TSH (UIU/mL) < 0.8 x LLN: number analyzed (Participants) | 8 | 10 | 8 | 10 | 11 | 29
  TSH (UIU/mL) < 0.8 x LLN | 0 | 2 | 0 | 0 | 1 | 4
  TSH (UIU/mL) > 1.2 x ULN: number analyzed (Participants) | 8 | 10 | 8 | 10 | 11 | 29
  TSH (UIU/mL) > 1.2 x ULN | 2 | 3 | 4 | 4 | 3 | 5
  Glucose (mg/dL) < 0.6 x LLN | 0 | 0 | 0 | 0 | 0 | 1
  Glucose (mg/dL) > 1.5 x ULN | 0 | 3 | 3 | 2 | 1 | 10
  Creatine Kinase (CK) (U/L) > 2.0 x ULN: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 1
  Creatine Kinase (CK) (U/L) > 2.0 x ULN |  |  |  | 0 |  | 0
  Amylase (U/L) > 1.5 x ULN | 2 | 1 | 2 | 0 | 0 | 3
  Lipase (U/L) > 1.5 x ULN | 1 | 3 | 2 | 0 | 0 | 7
  Urine Protein (Qual) >= 1 | 2 | 5 | 4 | 2 | 4 | 7
  Urine Blood/Hgb (Qual) >= 1: number analyzed (Participants) | 10 | 12 | 12 | 10 | 10 | 28
  Urine Blood/Hgb (Qual) >= 1 | 2 | 5 | 4 | 1 | 3 | 7
  Urine RBC (/HPF) >= 20: number analyzed (Participants) | 10 | 12 | 10 | 10 | 11 | 22
  Urine RBC (/HPF) >= 20 | 1 | 3 | 1 | 2 | 2 | 4
  Urine WBC (/HPF) >= 20: number analyzed (Participants) | 10 | 12 | 10 | 10 | 11 | 29
  Urine WBC (/HPF) >= 20 | 2 | 4 | 4 | 3 | 2 | 7
  Urine Epithelial Cells (/HPF) >= 6: number analyzed (Participants) | 8 | 10 | 9 | 7 | 6 | 12
  Urine Epithelial Cells (/HPF) >= 6 | 5 | 5 | 2 | 2 | 2 | 6
  Urine Casts (/LPF) > 1: number analyzed (Participants) | 5 | 3 | 3 | 3 | 3 | 12
  Urine Casts (/LPF) > 1 | 0 | 0 | 0 | 0 | 0 | 2
  Urine Granular Casts (/LPF) > 1: number analyzed (Participants) | 5 | 5 | 4 | 4 | 1 | 9
  Urine Granular Casts (/LPF) > 1 | 0 | 1 | 0 | 0 | 0 | 1
  Urine Hyaline Casts (/LPF) >1: number analyzed (Participants) | 5 | 7 | 5 | 5 | 5 | 11
  Urine Hyaline Casts (/LPF) >1 | 1 | 2 | 2 | 0 | 4 | 5
  Urine Bacteria (/HPF) > 20: number analyzed (Participants) | 7 | 10 | 10 | 9 | 10 | 18
  Urine Bacteria (/HPF) > 20 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Objective Response Rate (ORR) Assessed by Response Evaluation Criteria in Solid Tumor (RECIST) Version 1.1 and Immune Related Response Evaluation Criteria in Solid Tumors (irRECIST) in Part A
Description: ORR was defined as the percentage of patients with best overall response (BOR) of CR or PR relative to the appropriate analysis set.
  CR: Complete response is defined (per RECIST 1.1) as disappearance of all target and non target lesions. Any pathological lymph nodes (whether target or non target) must have reduction in short axis to <10 mm.
  PR: Partial response is difined (per RECIST 1.1) as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Overall immune related complete response (irCR): Complete disappearance of all lesions (whether measurable or not) and no new lesions. All measurable lymph nodes also must have a reduction in short axis to <10 mm.
  Overall immune related partial response (irPR): Sum of the diameters (longest for non nodal lesions, shortest for nodal lesions) of target and new measurable lesions decreases ≥30%.
Time Frame: Baseline up to 24 months post first dose.
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Part A1: PF-04518600 0.01mg/kg | Part A1: PF-04518600 0.1mg/kg | Part A1: PF-04518600 0.3mg/kg | Part A1: PF-04518600 1.5mg/kg | Part A1: PF-04518600 3.0mg/kg | Part A1: PF-04518600 10mg/kg | Part A2: PF-04518600 30mg | Part A2: PF-04518600 250mg
Number analyzed (Participants) | 2 | 10 | 11 | 12 | 13 | 4 | 16 | 19
percentage of participants
  ORR per RECIST v1.1 | 0 | 10 | 9.1 | 0 | 0 | 25 | 0 | 0
  ORR per irRECIST | 0 | 10 | 9.1 | 0 | 0 | 25 | 0 | 0

8. Secondary Outcome: Kaplan-Meier Estimate of Median Progression-Free Survival (PFS) in Part A
Description: PFS was defined as the time from randomization date to date of first documentation of progressive disease(PD) based on RECIST, irRECIST or death due to any cause.
  PD was progression documented after start date and not qualifying as CR, PR or SD per RECIST.
Time Frame: Baseline up to 24 months post first dose
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A1: PF-04518600 0.01mg/kg | Part A1: PF-04518600 0.1mg/kg | Part A1: PF-04518600 0.3mg/kg | Part A1: PF-04518600 1.5mg/kg | Part A1: PF-04518600 3.0mg/kg | Part A1: PF-04518600 10mg/kg | Part A2: PF-04518600 30mg | Part A2: PF-04518600 250mg
Number analyzed (Participants) | 2 | 10 | 11 | 12 | 13 | 4 | 16 | 19
months | 1.3 [1.3 to 1.4] | 3.5 [1.3 to 4.2] | 5.4 [1.3 to 24.0] | 1.4 [1.3 to 8.3] | 2.7 [1.3 to 5.6] | 4.8 [0.7 to NA] — The upper limit was not estimable. Because the upper limit for PFS based on Kaplan-Meier method was not reached. | 3.0 [1.5 to 3.7] | 2.8 [1.7 to 3.6]

9. Secondary Outcome: Kaplan-Meier Estimate of Median Time to Progression (TTP) in Part A
Description: TTP was defined as the time from start date to the date of the first documentation of PD. PD was documented after start date and not qualifying as CR, PR or SD per RECIST.
Time Frame: Baseline up to 24 months post first dose
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A1: PF-04518600 0.01mg/kg | Part A1: PF-04518600 0.1mg/kg | Part A1: PF-04518600 0.3mg/kg | Part A1: PF-04518600 1.5mg/kg | Part A1: PF-04518600 3.0mg/kg | Part A1: PF-04518600 10mg/kg | Part A2: PF-04518600 30mg | Part A2: PF-04518600 250mg
Number analyzed (Participants) | 2 | 10 | 11 | 12 | 13 | 4 | 16 | 19
months | 1.3 [1.3 to 1.4] | 4.1 [1.3 to 6.5] | 5.4 [1.3 to 24.0] | 1.4 [1.3 to 8.3] | 3.2 [1.2 to 5.6] | 8.3 [1.2 to NA] — The upper limit was not estimable. Because the upper limit for TTP based on Kaplan-Meier method was not reached. | 3.2 [1.5 to 3.7] | 2.8 [1.7 to 3.6]

10. Secondary Outcome: Number of Participants Having Stable Disease (SD) in Part A
Description: SD was defined as persistence of any non target lesions and/or tumor marker level above the normal limits.
Time Frame: Baseline up to 24 months post first dose.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part A1: PF-04518600 0.01mg/kg | Part A1: PF-04518600 0.1mg/kg | Part A1: PF-04518600 0.3mg/kg | Part A1: PF-04518600 1.5mg/kg | Part A1: PF-04518600 3.0mg/kg | Part A1: PF-04518600 10mg/kg | Part A2: PF-04518600 30mg | Part A2: PF-04518600 250mg
Number analyzed (Participants) | 2 | 10 | 11 | 12 | 13 | 4 | 16 | 19
Participants | 0 | 5 | 6 | 6 | 8 | 1 | 9 | 10

11. Secondary Outcome: Kaplan-Meier Estimate of Median Duration of Response (DoR) in Part A
Description: DoR was defined as the time from first documentation of PR or CR to date of first documentation of PD or death due to any cause for patients with an objective response.
  CR was defined as complete disappearance of all target lesions with the exception of nodal disease and all target nodes must decrease to normal size (short axis <10 mm) and all target lesions must be assessed.
  PR was defined as greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. The short diameter is used in the sum for target nodes, while the longest diameter is used in the sum for all other target lesions and all target lesions must be assessed.
Time Frame: Baseline up to 24 months post first dose.
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A1: PF-04518600 0.01mg/kg | Part A1: PF-04518600 0.1mg/kg | Part A1: PF-04518600 0.3mg/kg | Part A1: PF-04518600 1.5mg/kg | Part A1: PF-04518600 3.0mg/kg | Part A1: PF-04518600 10mg/kg | Part A2: PF-04518600 30mg | Part A2: PF-04518600 250mg
Number analyzed (Participants) | 2 | 10 | 11 | 12 | 13 | 4 | 16 | 19
months | NA [NA to NA] — Median value and ranges for 95% CI were not estimable due to no participants in this cohort achieved CR or PR. | 2.4 [NA to NA] — Ranges for 95% CI were not estimable due to less than 50% participants in this cohort achieved CR or PR. | 21.4 [NA to NA] — Ranges for 95% CI were not estimable due to less than 50% participants in this cohort achieved CR or PR. | NA [NA to NA] — Median value and ranges for 95% CI were not estimable due to no participants in this cohort achieved CR or PR. | NA [NA to NA] — Median value and ranges for 95% CI were not estimable due to no participants in this cohort achieved CR or PR. | NA [NA to NA] — Median value and ranges for 95% CI were not estimable due to no participants in this cohort achieved CR or PR. | NA [NA to NA] — Median value and ranges for 95% CI were not estimable due to no participants in this cohort achieved CR or PR. | NA [NA to NA] — Median value and ranges for 95% CI were not estimable due to no participants in this cohort achieved CR or PR.

12. Secondary Outcome: Kaplan-Meier Estimate of Median Overall Survival (OS) in Part A
Description: OS was defined as time in months from the start of study treatment to date of death due to any cause. OS was calculated as the death date or last known alive date (if death date unavailable) minus the date of first dose of study medication plus 1 divided by 30.44.
Time Frame: Baseline up to 24 months post first dose.
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A1: PF-04518600 0.01mg/kg | Part A1: PF-04518600 0.1mg/kg | Part A1: PF-04518600 0.3mg/kg | Part A1: PF-04518600 1.5mg/kg | Part A1: PF-04518600 3.0mg/kg | Part A1: PF-04518600 10mg/kg | Part A2: PF-04518600 30mg | Part A2: PF-04518600 250mg
Number analyzed (Participants) | 2 | 10 | 11 | 12 | 13 | 4 | 16 | 19
months | 11 [7.3 to 14.8] | 13.0 [3.3 to 20.7] | 17.6 [4.1 to NA] — The upper limit was not estimable. Because the upper limit for OS based on Kaplan-Meier method was not reached. | 9.0 [3.8 to 17.2] | 7.4 [5.1 to 19.1] | 7.5 [0.7 to NA] — The upper limit was not estimable. Because the upper limit for OS based on Kaplan-Meier method was not reached. | 15.6 [4.2 to NA] — The upper limit was not estimable. Because the upper limit for OS based on Kaplan-Meier method was not reached. | 23.9 [6.5 to NA] — The upper limit was not estimable. Because the upper limit for OS based on Kaplan-Meier method was not reached.

13. Secondary Outcome: Overall Survival Rates at Months 6, 12, and 24 in Part A
Description: Probability of survival at 6, 12, and 24 months after the first dose of study treatment.
Time Frame: Baseline up to 24 months post first dose.
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Probability of survival
Arm/Group | Part A1: PF-04518600 0.01mg/kg | Part A1: PF-04518600 0.1mg/kg | Part A1: PF-04518600 0.3mg/kg | Part A1: PF-04518600 1.5mg/kg | Part A1: PF-04518600 3.0mg/kg | Part A1: PF-04518600 10mg/kg | Part A2: PF-04518600 30mg | Part A2: PF-04518600 250mg
Number analyzed (Participants) | 2 | 10 | 11 | 12 | 13 | 4 | 16 | 19
Probability of survival
  Survival Probability at Month 6 | 100 [100 to 100] | 68.6 [30.5 to 88.7] | 88.9 [43.3 to 98.4] | 75.0 [40.8 to 91.2] | 67.7 [34.9 to 86.5] | 50.0 [5.8 to 84.5] | 62.5 [31.7 to 82.5] | 83.9 [57.9 to 94.5]
  Survival Probability at Month 12 | 50.0 [0.6 to 91.0] | 51.4 [14.3 to 79.6] | 55.6 [20.4 to 80.5] | 41.7 [15.2 to 66.5] | 33.8 [10.5 to 59.4] | 50.0 [5.8 to 84.5] | 54.7 [25.4 to 76.6] | 58.4 [31.6 to 77.8]
  Survival Probability at Month 24 | NA [NA to NA] — Number and ranges for 95% CI were not estimable due to both participants in the group have been censored or died before month 24. | NA [NA to NA] — Number and ranges for 95% CI were not estimable due to all participants in the group have been censored or died before month 24. | 44.4 [13.6 to 71.9] | NA [NA to NA] — Number and ranges for 95% CI were not estimable due to all participants in the group have been censored or died before month 24. | 16.9 [2.7 to 41.7] | 25.0 [0.9 to 66.5] | 27.3 [6.9 to 53.4] | 42.6 [17.7 to 65.7]

14. Secondary Outcome: Maximum Serum Concentration (Cmax) of PF-04518600 Following Single Dose on Cycle 1 Day 1 (C1D1) and Steady-State Maximum Serum Concentration(Css,Max) Following Multiple Doses on Cycle 3 Day 1 (C3D1) in Part A
Description: Cmax was defined as maximum observed serum concentration and can be observed directly from data.
  Css,max was the Cmax on C3D1.
Time Frame: For Part A1, pre-dose, 1, 4, and 24 hours post dose on C1D1, pre-dose, 1, and 4 hours post dose on Day 1 of Cycles 3; For Par A2, pre-dose, 1, and 4 hours post dose on C1D1, pre-dose and 1 hour post dose on Day 1 of Cycles 3.
Population: The pharmacokinetic (PK) parameter analysis population was defined as all enrolled participants treated who had sufficient information to estimate at least 1 of the PK parameters of interest. Number of participants analyzed represents the total number of participants in each treatment group in the PK parameter analysis population. Number analyzed represents the number of participants contributing to the summary statistics for Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (µg/mL)
Arm/Group | Part A1: PF-04518600 0.01mg/kg | Part A1: PF-04518600 0.1mg/kg | Part A1: PF-04518600 0.3mg/kg | Part A1: PF-04518600 1.5mg/kg | Part A1: PF-04518600 3.0mg/kg | Part A1: PF-04518600 10mg/kg | Part A2: PF-04518600 30mg | Part A2: PF-04518600 250mg
Number analyzed (Participants) | 1 | 10 | 10 | 12 | 13 | 4 | 16 | 19
microgram/milliliter (µg/mL)
  CYCLE1/DAY1 | 0.231 (NA) — Geometric CV was not calculated for n<3. | 2.871 (24) | 8.448 (17) | 36.71 (21) | 75.91 (18) | 268.1 (20) | 8.264 (25) | 72.05 (22)
  CYCLE3/DAY1: number analyzed (Participants) | 0 | 10 | 9 | 12 | 9 | 3 | 15 | 16
  CYCLE3/DAY1 |  | 2.731 (54) | 11.03 (23) | 56.15 (19) | 114.9 (22) | 401.1 (26) | 10.27 (32) | 105.7 (23)

15. Secondary Outcome: Area Under the Concentration-Time Profile From Time 0 to Time Tau (AUCtau) of PF-04518600 Following Single Dose on C1D1 and Following Multiple Doses on C3D1 in Part A
Description: AUCtau was defined as area under the concentration curve from time 0 to end of dosing interval where dosing interval was 2 weeks.
Time Frame: as for outcome 14
Population: The PK parameter analysis population was defined as all enrolled participants treated who had sufficient information to estimate at least 1 of the PK parameters of interest. Number of participants analyzed represents the total number of participants in each treatment group in the PK parameter analysis population. Number analyzed represents the number of participants contributing to the summary statistics for AUCtau.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram•hour/milliliter (µg•hr/mL)
Arm/Group | Part A1: PF-04518600 0.01mg/kg | Part A1: PF-04518600 0.1mg/kg | Part A1: PF-04518600 0.3mg/kg | Part A1: PF-04518600 1.5mg/kg | Part A1: PF-04518600 3.0mg/kg | Part A1: PF-04518600 10mg/kg | Part A2: PF-04518600 30mg | Part A2: PF-04518600 250mg
Number analyzed (Participants) | 1 | 10 | 10 | 12 | 13 | 4 | 16 | 19
microgram•hour/milliliter (µg•hr/mL)
  CYCLE1/DAY1: number analyzed (Participants) | 1 | 10 | 9 | 12 | 12 | 3 | 16 | 17
  CYCLE1/DAY1 | 7.59 (NA) — Geometric CV was not calculated for n<3. | 303.5 (35) | 1350 (20) | 6218 (23) | 12810 (17) | 38220 (19) | 1375 (25) | 14360 (19)
  CYCLE3/DAY1: number analyzed (Participants) | 0 | 8 | 7 | 7 | 8 | 3 | 14 | 15
  CYCLE3/DAY1 |  | 299 (151) | 2072 (36) | 11610 (18) | 25600 (21) | 82710 (32) | 2236 (37) | 25380 (29)

16. Secondary Outcome: Area Under the Concentration-Time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) of PF-04518600 Following Single Dose on C1D1 and Following Multiple Doses on C3D1 in Part A
Description: AUCinf was defined as area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). It was obtained from AUC (0-t) plus AUC (t-inf).
Time Frame: as for outcome 14
Population: The PK parameter analysis population was defined as all enrolled participants treated who had sufficient information to estimate at least 1 of the PK parameters of interest. Number of participants analyzed represents the total number of participants in each treatment group in the PK parameter analysis population. Number analyzed represents the number of participants contributing to the summary statistics for AUCinf.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*hr/mL
Arm/Group | Part A1: PF-04518600 0.01mg/kg | Part A1: PF-04518600 0.1mg/kg | Part A1: PF-04518600 0.3mg/kg | Part A1: PF-04518600 1.5mg/kg | Part A1: PF-04518600 3.0mg/kg | Part A1: PF-04518600 10mg/kg | Part A2: PF-04518600 30mg | Part A2: PF-04518600 250mg
Number analyzed (Participants) | 1 | 10 | 10 | 12 | 13 | 4 | 16 | 19
μg*hr/mL
  CYCLE1/DAY1: number analyzed (Participants) | 0 | 8 | 2 | 0 | 1 | 0 | 2 | 1
  CYCLE1/DAY1 |  | 293.7 (34) | NA (NA) — Geometric Mean and Geometric CV was not calculated for n<3. And the individual values were 1590,1010. |  | 23000 (NA) — Geometric CV was not calculated for n<3. |  | NA (NA) — Geometric Mean and Geometric CV was not calculated for n<3. And the individual values were 1580,991. | 22700 (NA) — Geometric CV was not calculated for n<3.
  CYCLE3/DAY1: number analyzed (Participants) | 0 | 5 | 0 | 0 | 1 | 0 | 1 | 1
  CYCLE3/DAY1 |  | 380.7 (56) |  |  | 33800 (NA) — Geometric CV was not calculated for n<3. |  | 1180 (NA) — Geometric CV was not calculated for n<3. | 35000 (NA) — Geometric CV was not calculated for n<3.

17. Secondary Outcome: Terminal Half-Life (t1/2) of PF-04518600 Following Single Dose on C1D1 and Following Multiple Doses on C3D1 in Part A
Description: t1/2 was defined as the time measured for the serum concentration to decrease by one half of the initial concentration.
Time Frame: as for outcome 14
Population: The PK parameter analysis population was defined as all enrolled participants treated who had sufficient information to estimate at least 1 of the PK parameters of interest. Number of participants analyzed represents the total number of participants in each treatment group in the PK parameter analysis population. Number analyzed represents the number of participants contributing to the summary statistics for t1/2.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Part A1: PF-04518600 0.01mg/kg | Part A1: PF-04518600 0.1mg/kg | Part A1: PF-04518600 0.3mg/kg | Part A1: PF-04518600 1.5mg/kg | Part A1: PF-04518600 3.0mg/kg | Part A1: PF-04518600 10mg/kg | Part A2: PF-04518600 30mg | Part A2: PF-04518600 250mg
Number analyzed (Participants) | 1 | 10 | 10 | 12 | 13 | 4 | 16 | 19
days
  CYCLE1/DAY1: number analyzed (Participants) | 0 | 8 | 2 | 0 | 1 | 0 | 2 | 1
  CYCLE1/DAY1 |  | 3.410 (1.0992) | NA (NA) — Geometric Mean and Geometric CV was not calculated for n<3. And the individual values were 5.77,4.83. |  | 13.1 (NA) — Geometric CV was not calculated for n<3. |  | 5.67 (5.89) | 11.9 (NA) — Geometric CV was not calculated for n<3.
  CYCLE3/DAY1: number analyzed (Participants) | 0 | 5 | 0 | 0 | 1 | 0 | 1 | 1
  CYCLE3/DAY1 |  | 4.010 (1.1370) |  |  | 10.6 (NA) — Geometric CV was not calculated for n<3. |  | 5.76 (NA) — Geometric CV was not calculated for n<3. | 11.9 (NA) — Geometric CV was not calculated for n<3.

18. Secondary Outcome: Lowest Serum Concentration Observed During the Dosing Interval (Cmin) of PF-04518600 Following Multiple Doses on C3D1 in Part A.
Description: Cmin was defined as Lowest concentration observed during the dosing interval and can be observed directly from data.
Time Frame: as for outcome 14
Population: The PK parameter analysis population was defined as all enrolled participants treated who had sufficient information to estimate at least 1 of the PK parameters of interest. Number of participants analyzed represents the total number of participants in each treatment group in the PK parameter analysis population. Number analyzed represents the number of participants contributing to the summary statistics for Cmin.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part A1: PF-04518600 0.01mg/kg | Part A1: PF-04518600 0.1mg/kg | Part A1: PF-04518600 0.3mg/kg | Part A1: PF-04518600 1.5mg/kg | Part A1: PF-04518600 3.0mg/kg | Part A1: PF-04518600 10mg/kg | Part A2: PF-04518600 30mg | Part A2: PF-04518600 250mg
Number analyzed (Participants) | 0 | 10 | 9 | 12 | 9 | 3 | 15 | 16
ug/mL |  | 0.05952 (51749) | 2.882 (61) | 17.79 (32) | 36.14 (48) | 130 (41) | 2.968 (55) | 37.62 (47)

19. Secondary Outcome: Average Serum Concentration Over the Dosing Interval (Cav) of PF-04518600 Following Multiple Doses on C3D1 in Part A
Description: Cav was defined as average serum concentration over the dosing interval.
Time Frame: as for outcome 14
Population: The PK parameter analysis population was defined as all enrolled participants treated who had sufficient information to estimate at least 1 of the PK parameters of interest. Number of participants analyzed represents the total number of participants in each treatment group in the PK parameter analysis population. Number analyzed represents the number of participants contributing to the summary statistics for Cav.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part A1: PF-04518600 0.01mg/kg | Part A1: PF-04518600 0.1mg/kg | Part A1: PF-04518600 0.3mg/kg | Part A1: PF-04518600 1.5mg/kg | Part A1: PF-04518600 3.0mg/kg | Part A1: PF-04518600 10mg/kg | Part A2: PF-04518600 30mg | Part A2: PF-04518600 250mg
Number analyzed (Participants) | 0 | 8 | 7 | 7 | 8 | 3 | 14 | 15
µg/mL |  | 0.8897 (151) | 6.166 (36) | 34.55 (18) | 76.13 (20) | 246.1 (32) | 6.659 (37) | 75.55 (29)

20. Secondary Outcome: Clearance (CL) of PF-04518600 Following Multiple Doses on C3D1 in Part A
Description: Drug clearance was a quantitative measure of the rate at which a drug substance is removed from the blood (rate at which a drug is metabolized or eliminated by normal biological processes). CL=Dose/AUCss,tau
Time Frame: as for outcome 14
Population: The PK parameter analysis population was defined as all enrolled participants treated who had sufficient information to estimate at least 1 of the PK parameters of interest. Number of participants analyzed represents the total number of participants in each treatment group in the PK parameter analysis population. Number analyzed represents the number of participants contributing to the summary statistics for CL.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter/hour/kilogram (mL/hr/kg)
Arm/Group | Part A1: PF-04518600 0.01mg/kg | Part A1: PF-04518600 0.1mg/kg | Part A1: PF-04518600 0.3mg/kg | Part A1: PF-04518600 1.5mg/kg | Part A1: PF-04518600 3.0mg/kg | Part A1: PF-04518600 10mg/kg | Part A2: PF-04518600 30mg | Part A2: PF-04518600 250mg
Number analyzed (Participants) | 0 | 8 | 7 | 7 | 8 | 3 | 14 | 15
milliliter/hour/kilogram (mL/hr/kg) |  | 0.3342 (151) | 0.1448 (48) | 0.1291 (18) | 0.1171 (21) | 0.1209 (32) | 0.1739 (28) | 0.1423 (31)

21. Secondary Outcome: Apparent Volume of Distribution at Steady State (Vss) of PF-04518600 Following Multiple Doses on C3D1 in Part A.
Description: Vss was defined as volume of distribution at steady state.
Time Frame: as for outcome 14
Population: The PK parameter analysis population was defined as all enrolled participants treated who had sufficient information to estimate at least 1 of the PK parameters of interest. Number of participants analyzed represents the total number of participants in each treatment group in the PK parameter analysis population. Number analyzed represents the number of participants contributing to the summary statistics for Vss.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter/kilograms (mL/kg)
Arm/Group | Part A1: PF-04518600 0.01mg/kg | Part A1: PF-04518600 0.1mg/kg | Part A1: PF-04518600 0.3mg/kg | Part A1: PF-04518600 1.5mg/kg | Part A1: PF-04518600 3.0mg/kg | Part A1: PF-04518600 10mg/kg | Part A2: PF-04518600 30mg | Part A2: PF-04518600 250mg
Number analyzed (Participants) | 0 | 5 | 0 | 0 | 1 | 0 | 1 | 1
milliliter/kilograms (mL/kg) |  | 39.17 (19) |  |  | 55.3 (NA) — Geometric CV was not calculated for n<3. |  | 79.2 (NA) — Geometric CV was not calculated for n<3. | 94.3 (NA) — Geometric CV was not calculated for n<3.

22. Secondary Outcome: Accumulation Ratio (Rac) of PF-04518600 at C3D1 Following Multiple Doses on C3D1 in Part A
Description: Accumulation ratio was calculated as, Rac obtained from Area Under the Concentration Time Curve (AUC) from Cycle 3 Day 1 divided by AUC from Cycle1 Day 1.
Time Frame: as for outcome 14
Population: The PK parameter analysis population was defined as all enrolled participants treated who had sufficient information to estimate at least 1 of the PK parameters of interest. Number of participants analyzed represents the total number of participants in each treatment group in the PK parameter analysis population. Number analyzed represents the number of participants contributing to the summary statistics for Rac.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part A1: PF-04518600 0.01mg/kg | Part A1: PF-04518600 0.1mg/kg | Part A1: PF-04518600 0.3mg/kg | Part A1: PF-04518600 1.5mg/kg | Part A1: PF-04518600 3.0mg/kg | Part A1: PF-04518600 10mg/kg | Part A2: PF-04518600 30mg | Part A2: PF-04518600 250mg
Number analyzed (Participants) | 0 | 8 | 6 | 7 | 8 | 3 | 14 | 15
ratio |  | 0.9893 (110) | 1.543 (32) | 1.785 (12) | 1.947 (12) | 2.161 (13) | 1.628 (19) | 1.709 (21)

23. Secondary Outcome: Number of Participants With Anti Drug Antibody (ADA) and Neutralizing Antibody (NAb) Against PF-04518600 in Part A
Description: ADA never-positive was defined as no positive ADA results at any time point. ADA ever-positive was defined as at least one positive ADA result at any time point. nAb never-positive was defined as no positive nAb results at any time point and nAb ever-positive was defined as at least one positive nAb result at any time point.
Time Frame: Baseline up to end of treatment (maximum of 14 weeks).
Population: The population included all enrolled participants with at least 1 of the ADA or NAb evaluated at pre- and/or post dose, and measurable PK concentrations.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A1: PF-04518600 0.01mg/kg | Part A1: PF-04518600 0.1mg/kg | Part A1: PF-04518600 0.3mg/kg | Part A1: PF-04518600 1.5mg/kg | Part A1: PF-04518600 3.0mg/kg | Part A1: PF-04518600 10mg/kg | Part A2: PF-04518600 30mg | Part A2: PF-04518600 250mg
Number analyzed (Participants) | 2 | 10 | 11 | 12 | 13 | 4 | 16 | 19
Participants
  ADA ever-positive: number analyzed (Participants) | 2 | 10 | 11 | 12 | 12 | 3 | 16 | 19
  ADA ever-positive | 2 | 9 | 5 | 2 | 0 | 0 | 7 | 0
  NAb ever-positive: number analyzed (Participants) | 2 | 10 | 11 | 12 | 12 | 3 | 16 | 19
  NAb ever-positive | 0 | 3 | 0 | 0 | 0 | 0 | 2 | 0

24. Secondary Outcome: Mean Unbound Cell Surface OX40 in Part A1
Description: Mean unbound cell surface OX40 in peripheral blood was measured to characterize the degree of target engagement (TE) by PF-04518600 at baseline and multiple doses.
Time Frame: Pre-dose, 4 and 24 hours post dose on Cycle 1 Day 1, and Day 8 on Cycles 1 to 3, then pre-dose on Cycles 4 and 7 and end of treatment in Part A1
Population: Analysis Population included all enrolled participants with at least 1 of the OX40 evaluated at pre and/or post dose.
Measure: Mean (Standard Deviation); unit: percentage of baseline concentration
Arm/Group | Part A1: PF-04518600 0.01mg/kg | Part A1: PF-04518600 0.1mg/kg | Part A1: PF-04518600 0.3mg/kg | Part A1: PF-04518600 1.5mg/kg | Part A1: PF-04518600 3.0mg/kg | Part A1: PF-04518600 10mg/kg
Number analyzed (Participants) | 2 | 8 | 10 | 9 | 8 | 4
percentage of baseline concentration
  Free, CD4+ Central Memory T Cells (%) Cycle 1 Day 1 (pre-dose): number analyzed (Participants) | 2 | 7 | 6 | 6 | 6 | 4
  Free, CD4+ Central Memory T Cells (%) Cycle 1 Day 1 (pre-dose) | 54.65 (15.203) | 51.54 (15.670) | 44.85 (9.407) | 41.53 (11.797) | 48.45 (18.597) | 47.60 (12.181)
  Free, CD4+ Central Memory T Cells (%) Cycle 1 Day 1 (4Hours(H)): number analyzed (Participants) | 2 | 7 | 6 | 5 | 6 | 4
  Free, CD4+ Central Memory T Cells (%) Cycle 1 Day 1 (4Hours(H)) | 33.60 (34.083) | 2.10 (2.621) | 0.53 (0.869) | 11.96 (26.576) | 0.40 (1.047) | -0.25 (0.507)
  Free, CD4+ Central Memory T Cells (%) Cycle 1 Day 2: number analyzed (Participants) | 2 | 7 | 6 | 7 | 7 | 2
  Free, CD4+ Central Memory T Cells (%) Cycle 1 Day 2 | 35.60 (31.961) | 2.19 (1.297) | 1.08 (0.859) | -0.07 (0.221) | 0.10 (0.469) | 0.10 (0.141)
  Free, CD4+ Central Memory T Cells (%) Cycle 1 Day 8: number analyzed (Participants) | 2 | 7 | 7 | 7 | 6 | 4
  Free, CD4+ Central Memory T Cells (%) Cycle 1 Day 8 | 53.90 (21.355) | 6.21 (6.127) | 0.94 (1.250) | 0.30 (0.306) | 0.70 (1.724) | -0.00 (0.294)
  Free, CD4+ Central Memory T Cells (%) Cycle 2 Day 1 (pre-dose): number analyzed (Participants) | 2 | 7 | 7 | 7 | 6 | 3
  Free, CD4+ Central Memory T Cells (%) Cycle 2 Day 1 (pre-dose) | 32.30 (11.738) | 15.21 (11.219) | 3.67 (2.511) | 0.41 (0.745) | 0.88 (1.881) | -0.03 (0.153)
  Free, CD4+ Central Memory T Cells (%) Cycle 2 Day 8: number analyzed (Participants) | 2 | 4 | 7 | 7 | 5 | 3
  Free, CD4+ Central Memory T Cells (%) Cycle 2 Day 8 | 46.35 (11.950) | 10.00 (6.387) | 1.26 (1.367) | 0.04 (0.098) | 0.24 (0.720) | -0.03 (0.058)
  Free, CD4+ Central Memory T Cells (%) Cycle 3 Day 1 (pre-dose): number analyzed (Participants) | 2 | 7 | 7 | 7 | 5 | 2
  Free, CD4+ Central Memory T Cells (%) Cycle 3 Day 1 (pre-dose) | 49.25 (21.708) | 27.44 (24.644) | 2.39 (3.102) | 0.04 (0.223) | 0.56 (0.940) | -0.20 (0.424)
  Free, CD4+ Central Memory T Cells (%) Cycle 3 Day 8: number analyzed (Participants) | 2 | 6 | 7 | 7 | 5 | 3
  Free, CD4+ Central Memory T Cells (%) Cycle 3 Day 8 | 35.15 (35.426) | 17.42 (18.026) | 1.03 (2.177) | 0.04 (0.151) | 0.44 (1.043) | -0.27 (0.379)
  Free, CD4+ Central Memory T Cells (%) Cycle 4 Day 1 (pre-dose): number analyzed (Participants) | 1 | 5 | 5 | 3 | 3 | 2
  Free, CD4+ Central Memory T Cells (%) Cycle 4 Day 1 (pre-dose) | 19.00 (NA) — There was only one participant with an assessment of free CD4+ central memory T cells on cycle 4 day 1 (pre-dose), therefore the deviation value was not calculated. | 22.54 (20.118) | 0.44 (0.391) | -0.07 (0.153) | 0.57 (1.069) | 0.20 (0.283)
  Free, CD4+ Central Memory T Cells (%) Cycle 7 Day 1 (pre-dose): number analyzed (Participants) | 0 | 4 | 3 | 1 | 3 | 2
  Free, CD4+ Central Memory T Cells (%) Cycle 7 Day 1 (pre-dose) |  | 24.3 (15.719) | 0.67 (0.603) | 0.10 (NA) — There was only one participant with an assessment of free CD4+ central memory T cells on cycle 7 day 1 (pre-dose), therefore the deviation value was not calculated. | 0.80 (1.386) | -0.25 (0.354)
  Free, CD4+ Central Memory T Cells (%) End of treatment: number analyzed (Participants) | 2 | 3 | 3 | 4 | 2 | 0
  Free, CD4+ Central Memory T Cells (%) End of treatment | 53.20 (1.838) | 31.13 (22.871) | 0.23 (0.252) | -0.18 (0.150) | 0.85 (1.061) |
  Free, CD4+ Effector Memory T Cells (%) Cycle 1 Day 1 (pre-dose): number analyzed (Participants) | 2 | 7 | 6 | 6 | 6 | 4
  Free, CD4+ Effector Memory T Cells (%) Cycle 1 Day 1 (pre-dose) | 66.95 (22.698) | 57.26 (18.236) | 55.18 (10.939) | 45.67 (12.565) | 42.72 (9.957) | 49.25 (15.295)
  Free, CD4+ Effector Memory T Cells (%) Cycle 1 Day 1 (4H): number analyzed (Participants) | 2 | 7 | 6 | 5 | 6 | 4
  Free, CD4+ Effector Memory T Cells (%) Cycle 1 Day 1 (4H) | 46.55 (41.366) | 3.41 (2.948) | 0.65 (0.771) | 12.92 (28.499) | 0.13 (0.333) | 0.08 (0.222)
  Free, CD4+ Effector Memory T Cells (%) Cycle 1 Day 2: number analyzed (Participants) | 2 | 7 | 6 | 7 | 7 | 2
  Free, CD4+ Effector Memory T Cells (%) Cycle 1 Day 2 | 44.35 (36.275) | 6.33 (5.863) | 2.70 (3.344) | 0.10 (0.238) | 0.01 (0.107) | -0.05 (0.071)
  Free, CD4+ Effector Memory T Cells (%) Cycle 1 Day 8: number analyzed (Participants) | 2 | 7 | 7 | 7 | 6 | 4
  Free, CD4+ Effector Memory T Cells (%) Cycle 1 Day 8 | 61.40 (21.072) | 11.50 (8.179) | 1.34 (1.646) | 0.66 (1.037) | 0.42 (0.624) | 0.08 (0.222)
  Free, CD4+ Effector Memory T Cells (%) Cycle 2 Day 1 (pre-dose): number analyzed (Participants) | 2 | 7 | 7 | 7 | 6 | 3
  Free, CD4+ Effector Memory T Cells (%) Cycle 2 Day 1 (pre-dose) | 51.55 (0.495) | 20.17 (12.575) | 4.83 (3.810) | 1.13 (1.908) | 0.58 (0.697) | -0.10 (0.173)
  Free, CD4+ Effector Memory T Cells (%) Cycle 2 Day 8: number analyzed (Participants) | 2 | 4 | 7 | 7 | 5 | 3
  Free, CD4+ Effector Memory T Cells (%) Cycle 2 Day 8 | 54.70 (20.648) | 19.42 (10.402) | 2.91 (2.195) | 0.23 (0.390) | 0.14 (0.385) | 0.30 (0.458)
  Free, CD4+ Effector Memory T Cells (%) Cycle 3 Day 1 (pre-dose): number analyzed (Participants) | 2 | 7 | 7 | 7 | 5 | 2
  Free, CD4+ Effector Memory T Cells (%) Cycle 3 Day 1 (pre-dose) | 60.20 (24.183) | 32.47 (23.479) | 3.49 (4.759) | 0.37 (0.556) | 0.16 (0.422) | -0.05 (0.071)
  Free, CD4+ Effector Memory T Cells (%) Cycle 3 Day 8: number analyzed (Participants) | 2 | 6 | 7 | 7 | 5 | 3
  Free, CD4+ Effector Memory T Cells (%) Cycle 3 Day 8 | 45.95 (41.083) | 24.00 (18.939) | 2.99 (4.632) | 0.11 (0.393) | 0.18 (0.349) | -0.03 (0.115)
  Free, CD4+ Effector Memory T Cells (%) Cycle 4 Day 1 (pre-dose): number analyzed (Participants) | 1 | 5 | 5 | 3 | 3 | 2
  Free, CD4+ Effector Memory T Cells (%) Cycle 4 Day 1 (pre-dose) | 21.10 (NA) — There was only one participant with an assessment of free CD4+ effector memory T cells on cycle 4 day 1 (pre-dose), therefore the deviation value was not calculated. | 24.52 (22.304) | 1.98 (1.096) | 0.13 (0.231) | 0.17 (0.289) | 0.15 (0.071)
  Free, CD4+ Effector Memory T Cells (%) Cycle 7 Day 1 (pre-dose): number analyzed (Participants) | 0 | 4 | 3 | 1 | 3 | 2
  Free, CD4+ Effector Memory T Cells (%) Cycle 7 Day 1 (pre-dose) |  | 32.88 (16.059) | 1.77 (1.966) | 0.00 (NA) — There was only one participant with an assessment of free CD4+ effector memory T cells on cycle 7 day 1 (pre-dose), therefore the deviation value was not calculated. | 0.37 (0.635) | -0.15 (0.071)
  Free, CD4+ Effector Memory T Cells (%) End of treatment: number analyzed (Participants) | 2 | 3 | 3 | 4 | 2 | 0
  Free, CD4+ Effector Memory T Cells (%) End of treatment | 58.05 (9.263) | 47.80 (21.140) | 0.27 (0.351) | 0.15 (0.436) | 0.50 (0.424) |
  Free, CD8+ Central Memory T Cells (%) Cycle 1 Day 1 (pre-dose): number analyzed (Participants) | 2 | 7 | 6 | 6 | 6 | 4
  Free, CD8+ Central Memory T Cells (%) Cycle 1 Day 1 (pre-dose) | 8.20 (0.566) | 9.77 (11.267) | 5.50 (4.018) | 12.52 (8.946) | 8.95 (6.649) | 18.73 (18.566)
  Free, CD8+ Central Memory T Cells (%) Cycle 1 Day 1 (4H): number analyzed (Participants) | 2 | 7 | 6 | 5 | 6 | 4
  Free, CD8+ Central Memory T Cells (%) Cycle 1 Day 1 (4H) | 3.40 (4.384) | 0.04 (0.730) | 0.65 (0.909) | 3.50 (7.275) | 1.13 (1.997) | 0.28 (0.457)
  Free, CD8+ Central Memory T Cells (%) Cycle 1 Day 2: number analyzed (Participants) | 2 | 7 | 6 | 7 | 7 | 2
  Free, CD8+ Central Memory T Cells (%) Cycle 1 Day 2 | 3.90 (1.273) | 0.59 (1.415) | 0.23 (0.674) | 0.03 (1.021) | 0.17 (0.836) | -0.20 (0.141)
  Free, CD8+ Central Memory T Cells (%) Cycle 1 Day 8: number analyzed (Participants) | 2 | 7 | 7 | 7 | 6 | 4
  Free, CD8+ Central Memory T Cells (%) Cycle 1 Day 8 | 3.20 (1.273) | 3.01 (4.378) | 0.54 (1.381) | -0.23 (0.699) | 1.13 (3.862) | -0.00 (0.408)
  Free, CD8+ Central Memory T Cells (%) Cycle 2 Day 1 (pre-dose): number analyzed (Participants) | 2 | 8 | 7 | 7 | 6 | 3
  Free, CD8+ Central Memory T Cells (%) Cycle 2 Day 1 (pre-dose) | 2.75 (3.465) | 3.91 (2.967) | 0.19 (0.937) | 0.31 (0.825) | 1.67 (4.089) | -0.20 (0.985)
  Free, CD8+ Central Memory T Cells (%) Cycle 2 Day 8: number analyzed (Participants) | 2 | 4 | 7 | 7 | 5 | 3
  Free, CD8+ Central Memory T Cells (%) Cycle 2 Day 8 | 4.50 (0.566) | 3.08 (2.994) | 0.31 (0.965) | -0.20 (0.673) | 1.20 (3.333) | 0.50 (0.600)
  Free, CD8+ Central Memory T Cells (%) Cycle 3 Day 1 (pre-dose): number analyzed (Participants) | 2 | 7 | 7 | 7 | 5 | 2
  Free, CD8+ Central Memory T Cells (%) Cycle 3 Day 1 (pre-dose) | 5.40 (5.091) | 6.81 (7.484) | 0.03 (0.699) | -0.26 (0.616) | 1.52 (3.702) | -0.40 (0.707)
  Free, CD8+ Central Memory T Cells (%) Cycle 3 Day 8: number analyzed (Participants) | 2 | 6 | 7 | 7 | 5 | 3
  Free, CD8+ Central Memory T Cells (%) Cycle 3 Day 8 | 3.00 (1.838) | 5.35 (4.214) | 0.53 (0.647) | -0.24 (1.086) | 0.44 (1.205) | -0.87 (0.681)
  Free, CD8+ Central Memory T Cells (%) Cycle 4 Day 1 (pre-dose): number analyzed (Participants) | 1 | 5 | 5 | 3 | 3 | 2
  Free, CD8+ Central Memory T Cells (%) Cycle 4 Day 1 (pre-dose) | 0.90 (NA) — There was only one participant with an assessment of free CD8+ central memory T cells on cycle 4 day 1 (pre-dose), therefore the deviation value was not calculated. | 5.06 (5.735) | -0.46 (1.561) | -0.03 (0.231) | 4.63 (8.372) | -0.45 (0.212)
  Free, CD8+ Central Memory T Cells (%) Cycle 7 Day 1 (pre-dose): number analyzed (Participants) | 0 | 4 | 3 | 1 | 3 | 2
  Free, CD8+ Central Memory T Cells (%) Cycle 7 Day 1 (pre-dose) |  | 6.55 (5.978) | 0.63 (1.274) | 0.40 (NA) — There was only one participant with an assessment of free CD8+ central memory T cells on cycle 7 day 1 (pre-dose), therefore the deviation value was not calculated. | 1.90 (3.897) | -0.60 (0.707)
  Free, CD8+ Central Memory T Cells (%) End of treatment: number analyzed (Participants) | 2 | 3 | 3 | 4 | 2 | 0
  Free, CD8+ Central Memory T Cells (%) End of treatment | 6.10 (6.647) | 9.80 (11.895) | -0.07 (0.115) | -0.27 (1.396) | 3.55 (5.445) |
  Free, CD8+ Effector Memory T Cells (%) Cycle 1 Day 1 (pre-dose): number analyzed (Participants) | 2 | 8 | 6 | 6 | 6 | 4
  Free, CD8+ Effector Memory T Cells (%) Cycle 1 Day 1 (pre-dose) | 2.55 (0.778) | 3.14 (2.932) | 2.05 (1.993) | 4.57 (2.953) | 3.15 (2.473) | 7.23 (8.066)
  Free, CD8+ Effector Memory T Cells (%) Cycle 1 Day 1 (4H): number analyzed (Participants) | 2 | 4 | 6 | 5 | 6 | 4
  Free, CD8+ Effector Memory T Cells (%) Cycle 1 Day 1 (4H) | 1.90 (0.849) | 0.06 (0.360) | 0.07 (0.216) | 1.40 (2.859) | 0.57 (1.537) | 0.08 (0.050)
  Free, CD8+ Effector Memory T Cells (%) Cycle 1 Day 2: number analyzed (Participants) | 2 | 7 | 6 | 7 | 7 | 2
  Free, CD8+ Effector Memory T Cells (%) Cycle 1 Day 2 | 1.05 (0.495) | 0.36 (0.519) | 0.05 (0.105) | 0.04 (0.151) | 0.41 (1.057) | -0.10 (0.000)
  Free, CD8+ Effector Memory T Cells (%) Cycle 1 Day 8: number analyzed (Participants) | 2 | 7 | 7 | 7 | 6 | 4
  Free, CD8+ Effector Memory T Cells (%) Cycle 1 Day 8 | 1.40 (0.283) | 0.50 (0.306) | -0.01 (0.146) | 0.03 (0.198) | 0.93 (2.647) | 0.00 (0.082)
  Free, CD8+ Effector Memory T Cells (%) Cycle 2 Day 1 (pre-dose): number analyzed (Participants) | 2 | 7 | 7 | 7 | 6 | 3
  Free, CD8+ Effector Memory T Cells (%) Cycle 2 Day 1 (pre-dose) | 1.85 (2.192) | 2.01 (2.507) | 0.04 (0.181) | 0.01 (0.090) | 1.37 (3.300) | 0.00 (0.100)
  Free, CD8+ Effector Memory T Cells (%) Cycle 2 Day 8: number analyzed (Participants) | 2 | 4 | 7 | 7 | 5 | 3
  Free, CD8+ Effector Memory T Cells (%) Cycle 2 Day 8 | 3.20 (2.404) | 1.10 (0.868) | 0.06 (0.172) | 0.06 (0.127) | 0.88 (2.080) | 0.07 (0.153)
  Free, CD8+ Effector Memory T Cells (%) Cycle 3 Day 1 (pre-dose): number analyzed (Participants) | 2 | 7 | 7 | 7 | 5 | 2
  Free, CD8+ Effector Memory T Cells (%) Cycle 3 Day 1 (pre-dose) | 2.75 (1.909) | 2.90 (2.725) | 0.17 (0.309) | -0.01 (0.135) | 0.32 (0.939) | -0.25 (0.212)
  Free, CD8+ Effector Memory T Cells (%) Cycle 3 Day 8: number analyzed (Participants) | 2 | 6 | 7 | 7 | 5 | 3
  Free, CD8+ Effector Memory T Cells (%) Cycle 3 Day 8 | 0.65 (0.636) | 2.50 (2.571) | 0.01 (0.107) | -0.06 (0.113) | 0.86 (1.596) | 0.00 (0.100)
  Free, CD8+ Effector Memory T Cells (%) Cycle 4 Day 1 (pre-dose): number analyzed (Participants) | 1 | 5 | 5 | 3 | 3 | 2
  Free, CD8+ Effector Memory T Cells (%) Cycle 4 Day 1 (pre-dose) | 2.20 (NA) — There was only one participant with an assessment of free CD8+ effector memory T cells on cycle 4 day 1 (pre-dose), therefore the deviation value was not calculated. | 3.06 (5.099) | 0.12 (0.164) | -0.07 (0.115) | 2.40 (4.244) | 0.15 (0.071)
  Free, CD8+ Effector Memory T Cells (%) Cycle 7 Day 1 (pre-dose): number analyzed (Participants) | 0 | 4 | 3 | 1 | 3 | 2
  Free, CD8+ Effector Memory T Cells (%) Cycle 7 Day 1 (pre-dose) |  | 4.28 (4.129) | 0.27 (0.462) | 0.20 (NA) — There was only one participant with an assessment of free CD8+ effector memory T cells on cycle 7 day 1 (pre-dose), therefore the deviation value was not calculated. | 1.13 (1.966) | -0.10 (0.000)
  Free, CD8+ Effector Memory T Cells (%) End of treatment: number analyzed (Participants) | 2 | 3 | 3 | 4 | 2 | 0
  Free, CD8+ Effector Memory T Cells (%) End of treatment | 2.05 (1.202) | 4.77 (7.218) | 0.30 (0.624) | -0.05 (0.058) | 1.00 (1.414) |
  Total, CD127lo Regulatory T Cells (%) Cycle 1 Day 1 (pre-dose): number analyzed (Participants) | 2 | 8 | 9 | 7 | 8 | 4
  Total, CD127lo Regulatory T Cells (%) Cycle 1 Day 1 (pre-dose) | 28.85 (0.778) | 40.18 (12.164) | 34.51 (10.649) | 42.13 (18.565) | 41.98 (12.160) | 38.35 (9.019)
  Total, CD127lo Regulatory T Cells (%) Cycle 1 Day 8: number analyzed (Participants) | 2 | 8 | 9 | 9 | 8 | 4
  Total, CD127lo Regulatory T Cells (%) Cycle 1 Day 8 | 26.85 (0.212) | 36.30 (10.886) | 34.46 (11.679) | 42.89 (13.179) | 40.23 (8.245) | 40.55 (9.219)
  Total, CD127lo Regulatory T Cells (%) Cycle 2 Day 1 (pre-dose): number analyzed (Participants) | 2 | 8 | 10 | 8 | 7 | 3
  Total, CD127lo Regulatory T Cells (%) Cycle 2 Day 1 (pre-dose) | 31.30 (1.980) | 35.28 (14.278) | 34.92 (5.867) | 40.88 (11.313) | 45.69 (6.950) | 38.43 (6.543)
  Total, CD127lo Regulatory T Cells (%) Cycle 2 Day 8: number analyzed (Participants) | 2 | 4 | 10 | 8 | 5 | 3
  Total, CD127lo Regulatory T Cells (%) Cycle 2 Day 8 | 27.55 (3.606) | 40.33 (15.040) | 38.21 (4.342) | 43.15 (9.439) | 52.44 (5.264) | 35.77 (14.935)
  Total, CD127lo Regulatory T Cells (%) Cycle 3 Day 1 (pre-dose): number analyzed (Participants) | 2 | 8 | 10 | 9 | 6 | 2
  Total, CD127lo Regulatory T Cells (%) Cycle 3 Day 1 (pre-dose) | 28.85 (2.758) | 39.14 (12.053) | 33.46 (11.820) | 37.88 (11.844) | 44.57 (13.038) | 39.25 (20.718)
  Total, CD127lo Regulatory T Cells (%) Cycle 3 Day 8: number analyzed (Participants) | 2 | 8 | 10 | 9 | 7 | 3
  Total, CD127lo Regulatory T Cells (%) Cycle 3 Day 8 | 30.40 (0.566) | 34.08 (8.806) | 32.47 (13.862) | 38.61 (13.391) | 41.61 (11.904) | 41.10 (15.125)
  Total, CD127lo Regulatory T Cells (%) Cycle 4 Day 1 (pre-dose): number analyzed (Participants) | 1 | 8 | 7 | 5 | 5 | 2
  Total, CD127lo Regulatory T Cells (%) Cycle 4 Day 1 (pre-dose) | 34.40 (NA) — There was only one participant with an assessment of total, CD127lo regulatory T cells on cycle 4 day 1 (pre-dose), therefore the deviation value was not calculated. | 36.50 (6.840) | 36.40 (4.627) | 32.20 (7.105) | 41.88 (12.275) | 35.85 (0.354)
  Total, CD127lo Regulatory T Cells (%) Cycle 7 Day 1 (pre-dose): number analyzed (Participants) | 0 | 5 | 4 | 2 | 3 | 2
  Total, CD127lo Regulatory T Cells (%) Cycle 7 Day 1 (pre-dose) |  | 38.64 (5.538) | 35.20 (3.350) | 25.70 (9.051) | 45.23 (9.955) | 48.25 (12.799)
  Total, CD127lo Regulatory T Cells (%) End of treatment: number analyzed (Participants) | 2 | 5 | 5 | 5 | 3 | 0
  Total, CD127lo Regulatory T Cells (%) End of treatment | 35.30 (2.404) | 34.00 (16.913) | 28.12 (16.961) | 38.10 (10.006) | 45.20 (10.611) |
  Total, CD4+ Central Memory T Cells (%) Cycle 1 Day 1 (pre-dose): number analyzed (Participants) | 2 | 7 | 6 | 6 | 6 | 4
  Total, CD4+ Central Memory T Cells (%) Cycle 1 Day 1 (pre-dose) | 49.90 (3.536) | 50.61 (16.877) | 44.38 (9.798) | 45.35 (13.300) | 52.28 (16.746) | 33.23 (16.607)
  Total, CD4+ Central Memory T Cells (%) Cycle 1 Day 1 (4H): number analyzed (Participants) | 2 | 7 | 6 | 5 | 6 | 4
  Total, CD4+ Central Memory T Cells (%) Cycle 1 Day 1 (4H) | 56.45 (6.010) | 52.19 (16.212) | 48.00 (14.287) | 51.86 (10.272) | 44.77 (24.667) | 36.05 (16.733)
  Total, CD4+ Central Memory T Cells (%) Cycle 1 Day 2: number analyzed (Participants) | 2 | 7 | 6 | 7 | 7 | 2
  Total, CD4+ Central Memory T Cells (%) Cycle 1 Day 2 | 52.85 (11.384) | 52.74 (14.199) | 48.67 (8.943) | 39.77 (12.347) | 45.11 (21.747) | 21.00 (4.101)
  Total, CD4+ Central Memory T Cells (%) Cycle 1 Day 8: number analyzed (Participants) | 2 | 7 | 7 | 7 | 6 | 4
  Total, CD4+ Central Memory T Cells (%) Cycle 1 Day 8 | 49.75 (18.880) | 46.47 (14.885) | 39.07 (13.011) | 45.09 (10.489) | 38.22 (20.166) | 27.70 (13.124)
  Total, CD4+ Central Memory T Cells (%) Cycle 2 Day 1 (pre-dose): number analyzed (Participants) | 2 | 7 | 7 | 7 | 8 | 3
  Total, CD4+ Central Memory T Cells (%) Cycle 2 Day 1 (pre-dose) | 49.90 (9.758) | 41.43 (14.750) | 41.21 (9.855) | 45.70 (10.567) | 45.17 (16.509) | 23.30 (11.811)
  Total, CD4+ Central Memory T Cells (%) Cycle 2 Day 8: number analyzed (Participants) | 2 | 4 | 7 | 7 | 5 | 3
  Total, CD4+ Central Memory T Cells (%) Cycle 2 Day 8 | 50.85 (8.132) | 49.08 (20.277) | 46.00 (7.485) | 41.00 (12.981) | 34.40 (17.363) | 23.27 (26.999)
  Total, CD4+ Central Memory T Cells (%) Cycle 3 Day 1 (pre-dose): number analyzed (Participants) | 2 | 7 | 7 | 7 | 5 | 2
  Total, CD4+ Central Memory T Cells (%) Cycle 3 Day 1 (pre-dose) | 49.75 (13.223) | 50.04 (13.227) | 40.76 (18.801) | 42.94 (11.357) | 37.22 (19.773) | 35.65 (31.183)
  Total, CD4+ Central Memory T Cells (%) Cycle 3 Day 8: number analyzed (Participants) | 2 | 6 | 7 | 7 | 5 | 3
  Total, CD4+ Central Memory T Cells (%) Cycle 3 Day 8 | 54.95 (8.839) | 45.20 (16.005) | 41.20 (20.054) | 42.87 (10.049) | 39.30 (13.509) | 37.37 (16.783)
  Total, CD4+ Central Memory T Cells (%) Cycle 4 Day 1 (pre-dose): number analyzed (Participants) | 2 | 5 | 5 | 3 | 3 | 2
  Total, CD4+ Central Memory T Cells (%) Cycle 4 Day 1 (pre-dose) | 37.20 (NA) — There was only one participant with an assessment of total CD4+ central memory T cells on cycle 4 day 1 (pre-dose), therefore the deviation value was not calculated. | 47.52 (15.688) | 41.42 (11.115) | 43.43 (5.788) | 30.37 (15.309) | 32.15 (19.304)
  Total, CD4+ Central Memory T Cells (%) Cycle 7 Day 1 (pre-dose): number analyzed (Participants) | 0 | 4 | 3 | 1 | 3 | 2
  Total, CD4+ Central Memory T Cells (%) Cycle 7 Day 1 (pre-dose) |  | 53.80 (9.098) | 36.67 (2.589) | 39.90 (NA) — There was only one participant with an assessment of total CD4+ central memory T cells on cycle 7 day 1 (pre-dose), therefore the deviation value was not calculated. | 27.27 (23.200) | 49.00 (27.294)
  Total, CD4+ Central Memory T Cells (%) End of treatment: number analyzed (Participants) | 2 | 3 | 3 | 4 | 2 | 0
  Total, CD4+ Central Memory T Cells (%) End of treatment | 52.75 (13.789) | 46.70 (12.775) | 24.80 (23.435) | 41.38 (6.111) | 34.65 (11.526) |
  Total, CD4+ Effector Memory T Cells (%) Cycle 1 Day 1 (pre-dose): number analyzed (Participants) | 2 | 7 | 6 | 6 | 6 | 4
  Total, CD4+ Effector Memory T Cells (%) Cycle 1 Day 1 (pre-dose) | 59.60 (16.546) | 56.10 (15.093) | 43.38 (23.693) | 47.03 (13.816) | 40.25 (12.277) | 41.58 (15.879)
  Total, CD4+ Effector Memory T Cells (%) Cycle 1 Day 1 (4H): number analyzed (Participants) | 2 | 7 | 6 | 5 | 6 | 4
  Total, CD4+ Effector Memory T Cells (%) Cycle 1 Day 1 (4H) | 60.65 (17.607) | 58.76 (16.535) | 50.53 (13.385) | 47.82 (15.437) | 31.28 (15.021) | 38.68 (19.538)
  Total, CD4+ Effector Memory T Cells (%) Cycle 1 Day 2: number analyzed (Participants) | 2 | 8 | 6 | 7 | 7 | 2
  Total, CD4+ Effector Memory T Cells (%) Cycle 1 Day 2 | 57.00 (19.658) | 59.39 (15.181) | 52.93 (9.347) | 37.09 (14.705) | 31.91 (17.122) | 24.25 (19.728)
  Total, CD4+ Effector Memory T Cells (%) Cycle 1 Day 8: number analyzed (Participants) | 2 | 7 | 7 | 7 | 6 | 4
  Total, CD4+ Effector Memory T Cells (%) Cycle 1 Day 8 | 56.20 (18.526) | 50.57 (12.243) | 45.09 (11.917) | 44.00 (13.558) | 31.87 (18.013) | 33.43 (10.754)
  Total, CD4+ Effector Memory T Cells (%) Cycle 2 Day 1 (pre-dose): number analyzed (Participants) | 2 | 7 | 7 | 7 | 6 | 3
  Total, CD4+ Effector Memory T Cells (%) Cycle 2 Day 1 (pre-dose) | 58.45 (18.173) | 49.54 (12.391) | 51.86 (9.906) | 44.06 (12.694) | 35.20 (14.024) | 30.40 (12.382)
  Total, CD4+ Effector Memory T Cells (%) Cycle 2 Day 8: number analyzed (Participants) | 2 | 4 | 7 | 7 | 5 | 3
  Total, CD4+ Effector Memory T Cells (%) Cycle 2 Day 8 | 56.40 (15.274) | 62.78 (19.629) | 51.01 (14.110) | 43.93 (14.824) | 33.48 (21.662) | 31.60 (21.458)
  Total, CD4+ Effector Memory T Cells (%) Cycle 3 Day 1 (pre-dose): number analyzed (Participants) | 2 | 7 | 7 | 7 | 5 | 2
  Total, CD4+ Effector Memory T Cells (%) Cycle 3 Day 1 (pre-dose) | 56.50 (18.526) | 56.11 (14.652) | 46.63 (22.926) | 43.71 (14.276) | 35.08 (19.484) | 42.35 (21.708)
  Total, CD4+ Effector Memory T Cells (%) Cycle 3 Day 8: number analyzed (Participants) | 2 | 6 | 7 | 7 | 5 | 3
  Total, CD4+ Effector Memory T Cells (%) Cycle 3 Day 8 | 60.85 (15.344) | 51.48 (21.069) | 45.60 (23.497) | 42.40 (13.966) | 41.88 (16.112) | 31.67 (18.151)
  Total, CD4+ Effector Memory T Cells (%) Cycle 4 Day 1 (pre-dose): number analyzed (Participants) | 1 | 5 | 5 | 3 | 3 | 2
  Total, CD4+ Effector Memory T Cells (%) Cycle 4 Day 1 (pre-dose) | 44.00 (NA) — There was only one participant with an assessment of total CD4+ effector memory T cells on cycle 4 day 1 (pre-dose), therefore the deviation value was not calculated. | 49.92 (11.834) | 48.54 (14.165) | 51.03 (10.119) | 29.60 (7.754) | 33.40 (30.830)
  Total, CD4+ Effector Memory T Cells (%) Cycle 7 Day 1 (pre-dose): number analyzed (Participants) | 0 | 4 | 3 | 1 | 3 | 2
  Total, CD4+ Effector Memory T Cells (%) Cycle 7 Day 1 (pre-dose) |  | 55.98 (10.071) | 38.67 (12.438) | 44.80 (NA) — There was only one participant with an assessment of total CD4+ effector memory T cells on cycle 7 day 1 (pre-dose), therefore the deviation value was not calculated. | 22.10 (18.857) | 59.75 (12.092)
  Total, CD4+ Effector Memory T Cells (%) End of treatment: number analyzed (Participants) | 2 | 3 | 3 | 4 | 2 | 0
  Total, CD4+ Effector Memory T Cells (%) End of treatment | 62.50 (20.789) | 63.00 (21.165) | 21.43 (17.010) | 29.83 (12.258) | 36.80 (12.869) |
  Total, CD8+ Central Memory T Cells (%) Cycle 1 Day 1 (pre-dose): number analyzed (Participants) | 2 | 7 | 6 | 6 | 6 | 4
  Total, CD8+ Central Memory T Cells (%) Cycle 1 Day 1 (pre-dose) | 7.55 (4.879) | 12.00 (10.795) | 9.02 (5.270) | 16.30 (11.546) | 12.82 (4.961) | 15.63 (20.503)
  Total, CD8+ Central Memory T Cells (%) Cycle 1 Day 1 (4H): number analyzed (Participants) | 2 | 7 | 6 | 5 | 6 | 4
  Total, CD8+ Central Memory T Cells (%) Cycle 1 Day 1 (4H) | 10.35 (6.859) | 11.34 (11.046) | 9.00 (5.355) | 18.72 (14.591) | 10.03 (8.477) | 15.23 (15.784)
  Total, CD8+ Central Memory T Cells (%) Cycle 1 Day 2: number analyzed (Participants) | 2 | 7 | 6 | 7 | 7 | 2
  Total, CD8+ Central Memory T Cells (%) Cycle 1 Day 2 | 7.30 (5.940) | 10.33 (9.138) | 8.65 (6.783) | 12.27 (10.298) | 11.93 (8.826) | 23.95 (34.295)
  Total, CD8+ Central Memory T Cells (%) Cycle 1 Day 8: number analyzed (Participants) | 2 | 8 | 7 | 7 | 6 | 4
  Total, CD8+ Central Memory T Cells (%) Cycle 1 Day 8 | 4.50 (1.131) | 9.53 (7.607) | 9.03 (10.168) | 15.81 (9.926) | 9.55 (7.987) | 10.65 (15.910)
  Total, CD8+ Central Memory T Cells (%) Cycle 2 Day 1 (pre-dose): number analyzed (Participants) | 2 | 7 | 7 | 7 | 6 | 3
  Total, CD8+ Central Memory T Cells (%) Cycle 2 Day 1 (pre-dose) | 8.70 (7.495) | 9.56 (10.163) | 9.50 (12.278) | 14.83 (11.588) | 10.42 (7.695) | 2.67 (1.570)
  Total, CD8+ Central Memory T Cells (%) Cycle 2 Day 8: number analyzed (Participants) | 2 | 4 | 7 | 7 | 5 | 3
  Total, CD8+ Central Memory T Cells (%) Cycle 2 Day 8 | 8.70 (5.798) | 12.13 (11.505) | 10.19 (13.521) | 12.89 (8.212) | 10.38 (10.295) | 2.77 (3.109)
  Total, CD8+ Central Memory T Cells (%) Cycle 3 Day 1 (pre-dose): number analyzed (Participants) | 2 | 7 | 7 | 7 | 5 | 2
  Total, CD8+ Central Memory T Cells (%) Cycle 3 Day 1 (pre-dose) | 6.05 (4.738) | 12.11 (7.990) | 10.49 (11.153) | 14.19 (9.905) | 9.86 (9.571) | 6.20 (4.525)
  Total, CD8+ Central Memory T Cells (%) Cycle 3 Day 8: number analyzed (Participants) | 2 | 6 | 7 | 7 | 5 | 3
  Total, CD8+ Central Memory T Cells (%) Cycle 3 Day 8 | 6.05 (1.626) | 11.55 (8.232) | 11.29 (13.434) | 13.90 (8.309) | 10.34 (8.769) | 3.00 (1.900)
  Total, CD8+ Central Memory T Cells (%) Cycle 4 Day 1 (pre-dose): number analyzed (Participants) | 1 | 5 | 5 | 3 | 3 | 2
  Total, CD8+ Central Memory T Cells (%) Cycle 4 Day 1 (pre-dose) | 5.90 (NA) — There was only one participant with an assessment of total CD8+ central memory T cells on cycle 4 day 1 (pre-dose), therefore the deviation value was not be calculated. | 11.54 (10.077) | 13.42 (8.546) | 13.60 (10.942) | 12.07 (12.360) | 4.75 (3.041)
  Total, CD8+ Central Memory T Cells (%) Cycle 7 Day 1 (pre-dose): number analyzed (Participants) | 0 | 4 | 3 | 1 | 3 | 2
  Total, CD8+ Central Memory T Cells (%) Cycle 7 Day 1 (pre-dose) |  | 16.35 (10.850) | 8.03 (1.528) | 21.60 (NA) — There was only one participant with an assessment of total CD8+ central memory T cells on cycle 7 day 1 (pre-dose), therefore the deviation valuewas not calculated. | 11.97 (12.051) | 6.30 (2.263)
  Total, CD8+ Central Memory T Cells (%) End of treatment: number analyzed (Participants) | 2 | 3 | 3 | 4 | 2 | 0
  Total, CD8+ Central Memory T Cells (%) End of treatment | 6.85 (3.182) | 13.77 (10.845) | 3.87 (5.065) | 15.08 (12.687) | 9.90 (13.576) |
  Total, CD8+ Effector Memory T Cells (%) Cycle 1 Day 1 (pre-dose): number analyzed (Participants) | 2 | 7 | 6 | 6 | 6 | 4
  Total, CD8+ Effector Memory T Cells (%) Cycle 1 Day 1 (pre-dose) | 3.35 (2.051) | 3.66 (3.062) | 3.25 (2.091) | 5.35 (4.700) | 3.82 (3.207) | 24.48 (26.779)
  Total, CD8+ Effector Memory T Cells (%) Cycle 1 Day 1 (4H): number analyzed (Participants) | 2 | 7 | 6 | 5 | 6 | 4
  Total, CD8+ Effector Memory T Cells (%) Cycle 1 Day 1 (4H) | 3.80 (1.697) | 4.31 (3.611) | 2.67 (2.081) | 4.86 (5.229) | 2.80 (3.454) | 22.53 (26.873)
  Total, CD8+ Effector Memory T Cells (%) Cycle 1 Day 2: number analyzed (Participants) | 2 | 7 | 6 | 7 | 7 | 2
  Total, CD8+ Effector Memory T Cells (%) Cycle 1 Day 2 | 2.60 (0.990) | 5.19 (3.873) | 2.73 (2.004) | 3.57 (4.130) | 3.14 (3.347) | 11.70 (15.839)
  Total, CD8+ Effector Memory T Cells (%) Cycle 1 Day 8: number analyzed (Participants) | 2 | 7 | 7 | 7 | 6 | 4
  Total, CD8+ Effector Memory T Cells (%) Cycle 1 Day 8 | 2.60 (1.273) | 3.54 (2.463) | 3.36 (5.108) | 4.50 (4.727) | 2.57 (3.222) | 17.88 (20.990)
  Total, CD8+ Effector Memory T Cells (%) Cycle 2 Day 1 (pre-dose): number analyzed (Participants) | 2 | 7 | 7 | 7 | 6 | 3
  Total, CD8+ Effector Memory T Cells (%) Cycle 2 Day 1 (pre-dose) | 3.25 (2.616) | 4.70 (4.031) | 3.77 (6.125) | 4.53 (4.511) | 3.12 (3.539) | 13.10 (19.341)
  Total, CD8+ Effector Memory T Cells (%) Cycle 2 Day 8: number analyzed (Participants) | 2 | 4 | 7 | 7 | 5 | 3
  Total, CD8+ Effector Memory T Cells (%) Cycle 2 Day 8 | 2.65 (0.778) | 3.90 (3.524) | 3.56 (5.524) | 4.06 (4.008) | 4.16 (5.786) | 19.07 (30.641)
  Total, CD8+ Effector Memory T Cells (%) Cycle 3 Day 1 (pre-dose): number analyzed (Participants) | 2 | 7 | 7 | 7 | 5 | 2
  Total, CD8+ Effector Memory T Cells (%) Cycle 3 Day 1 (pre-dose) | 2.50 (1.697) | 5.14 (4.446) | 3.69 (5.607) | 4.33 (3.693) | 3.14 (3.884) | 30.45 (38.537)
  Total, CD8+ Effector Memory T Cells (%) Cycle 3 Day 8: number analyzed (Participants) | 2 | 6 | 7 | 7 | 5 | 3
  Total, CD8+ Effector Memory T Cells (%) Cycle 3 Day 8 | 2.70 (0.990) | 4.48 (4.388) | 3.50 (5.568) | 4.57 (4.340) | 3.64 (3.832) | 18.67 (27.050)
  Total, CD8+ Effector Memory T Cells (%) Cycle 4 Day 1 (pre-dose): number analyzed (Participants) | 1 | 5 | 5 | 3 | 3 | 2
  Total, CD8+ Effector Memory T Cells (%) Cycle 4 Day 1 (pre-dose) | 3.00 (NA) — There was only one participant with an assessment of total CD8+ effector memory T cells on cycle 4 day 1 (pre-dose), therefore the deviation value was not calculated. | 4.66 (5.283) | 5.94 (5.734) | 8.23 (4.900) | 3.33 (5.024) | 2.60 (0.990)
  Total, CD8+ Effector Memory T Cells (%) Cycle 7 Day 1 (pre-dose): number analyzed (Participants) | 0 | 4 | 3 | 1 | 3 | 2
  Total, CD8+ Effector Memory T Cells (%) Cycle 7 Day 1 (pre-dose) |  | 6.18 (4.811) | 2.60 (1.952) | 7.80 (NA) — There was only one participant with an assessment of total CD8+ effector memory T cells on cycle 7 day 1 (pre-dose), therefore the deviation value was not calculated. | 3.67 (5.755) | 35.40 (46.528)
  Total, CD8+ Effector Memory T Cells (%) End of treatment: number analyzed (Participants) | 2 | 3 | 3 | 4 | 2 | 0
  Total, CD8+ Effector Memory T Cells (%) End of treatment | 1.70 (0.141) | 3.93 (4.957) | 0.57 (0.306) | 1.95 (1.605) | 1.25 (1.061) |
  Total, FOXP3+ Regulatory T Cells (%) Cycle 1 Day 1 (pre-dose): number analyzed (Participants) | 2 | 8 | 9 | 7 | 8 | 4
  Total, FOXP3+ Regulatory T Cells (%) Cycle 1 Day 1 (pre-dose) | 34.10 (0.283) | 40.98 (10.428) | 38.67 (8.521) | 41.20 (16.148) | 46.55 (10.978) | 41.18 (8.761)
  Total, FOXP3+ Regulatory T Cells (%) Cycle 1 Day 8: number analyzed (Participants) | 2 | 8 | 9 | 9 | 8 | 4
  Total, FOXP3+ Regulatory T Cells (%) Cycle 1 Day 8 | 27.15 (4.172) | 39.53 (7.635) | 37.20 (8.902) | 44.29 (11.058) | 44.80 (7.508) | 42.40 (7.165)
  Total, FOXP3+ Regulatory T Cells (%) Cycle 2 Day 1 (pre-dose): number analyzed (Participants) | 2 | 8 | 10 | 8 | 7 | 3
  Total, FOXP3+ Regulatory T Cells (%) Cycle 2 Day 1 (pre-dose) | 35.70 (5.940) | 42.29 (13.590) | 36.97 (7.219) | 45.23 (11.181) | 49.74 (10.086) | 40.57 (3.415)
  Total, FOXP3+ Regulatory T Cells (%) Cycle 2 Day 8: number analyzed (Participants) | 2 | 4 | 10 | 8 | 5 | 3
  Total, FOXP3+ Regulatory T Cells (%) Cycle 2 Day 8 | 30.95 (3.465) | 44.45 (14.962) | 40.53 (6.707) | 46.71 (10.444) | 56.66 (12.388) | 39.93 (16.671)
  Total, FOXP3+ Regulatory T Cells (%) Cycle 3 Day 1 (pre-dose): number analyzed (Participants) | 2 | 8 | 10 | 9 | 6 | 2
  Total, FOXP3+ Regulatory T Cells (%) Cycle 3 Day 1 (pre-dose) | 31.50 (9.051) | 42.69 (14.259) | 35.62 (13.117) | 42.36 (9.707) | 50.30 (10.907) | 46.75 (19.728)
  Total, FOXP3+ Regulatory T Cells (%) Cycle 3 Day 8: number analyzed (Participants) | 2 | 8 | 10 | 9 | 7 | 3
  Total, FOXP3+ Regulatory T Cells (%) Cycle 3 Day 8 | 34.30 (3.536) | 38.83 (8.536) | 35.78 (13.922) | 41.69 (10.489) | 47.16 (13.427) | 41.70 (13.089)
  Total, FOXP3+ Regulatory T Cells (%) Cycle 4 Day 1 (pre-dose): number analyzed (Participants) | 1 | 8 | 7 | 5 | 5 | 2
  Total, FOXP3+ Regulatory T Cells (%) Cycle 4 Day 1 (pre-dose) | 35.30 (NA) — There was only one participant with an assessment of total FOXP3+ regulatory T cells on cycle 4 day 1 (pre-dose), therefore the deviation value was not calculated. | 38.83 (8.658) | 41.89 (10.092) | 35.78 (10.316) | 46.00 (11.665) | 55.70 (14.001)
  Total, FOXP3+ Regulatory T Cells (%) Cycle 7 Day 1 (pre-dose): number analyzed (Participants) | 0 | 5 | 4 | 2 | 3 | 2
  Total, FOXP3+ Regulatory T Cells (%) Cycle 7 Day 1 (pre-dose) |  | 41.80 (3.149) | 41.23 (6.725) | 28.70 (0.849) | 43.40 (5.145) | 52.35 (15.344)
  Total, FOXP3+ Regulatory T Cells (%) End of treatment: number analyzed (Participants) | 2 | 5 | 5 | 5 | 3 | 0
  Total, FOXP3+ Regulatory T Cells (%) End of treatment | 38.50 (3.960) | 37.88 (15.626) | 35.60 (19.987) | 43.94 (10.685) | 48.57 (7.596) |

25. Secondary Outcome: ORR Assessed by RECIST Version 1.1 and irRECIST in Part B
Description: as for outcome 7
Time Frame: Baseline up to 24 months post first dose.
Population: Analysis population included all enrolled participants who received at least 1 full or partial IV infusion of study drug PF-04518600 and PF-05082566.
Measure: Number; unit: Percentage of participants
Arm/Group | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg | Part B2: PF-04518600 30mg + PF-05082566 20mg
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 11 | 30
Percentage of participants
  ORR per RECIST v1.1 | 0 | 8.3 | 8.3 | 0 | 0 | 3.3
  ORR per irRECIST | 0 | 8.3 | 8.3 | 0 | 0 | 3.3

26. Secondary Outcome: Kaplan-Meier Estimate of Median PFS in Part B
Description: as for outcome 8
Time Frame: Baseline up to 24 months post first dose.
Population: as for outcome 25
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg | Part B2: PF-04518600 30mg + PF-05082566 20mg
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 11 | 30
months | 1.4 [0.6 to 2.7] | 2.8 [0.9 to 4.2] | 2.3 [1.4 to 5.5] | 1.4 [1.2 to 2.7] | 1.4 [1.0 to 2.8] | 3.2 [1.7 to 3.7]

27. Secondary Outcome: Kaplan-Meier Estimate of Median TTP in Part B
Description: as for outcome 9
Time Frame: Baseline up to 24 months post first dose.
Population: as for outcome 25
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg | Part B2: PF-04518600 30mg + PF-05082566 20mg
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 11 | 30
months | 1.4 [0.6 to 2.7] | 2.8 [0.9 to 4.2] | 2.6 [1.4 to 5.5] | 1.4 [0.9 to 2.7] | 1.4 [1.0 to 2.8] | 3.3 [1.7 to 4.3]

28. Secondary Outcome: Number of Participants Having SD in Part B
Description: SD was defined as persistence of any non target lesions and/or tumor marker level above the normal limits.
Time Frame: Baseline up to 24 months post first dose.
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg | Part B2: PF-04518600 30mg + PF-05082566 20mg
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 11 | 30
Participants | 2 | 5 | 4 | 4 | 3 | 14

29. Secondary Outcome: Kaplan-Meier Estimate of Median DoR in Part B
Description: as for outcome 11
Time Frame: Baseline up to 24 months post first dose.
Population: as for outcome 25
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg | Part B2: PF-04518600 30mg + PF-05082566 20mg
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 11 | 30
months | NA [NA to NA] — Median and ranges for 95% CI were not estimable due to no participants in this cohort achieved CR or PR. | NA [NA to NA] — Median and ranges for 95% CI were not estimable due to no participants in this cohort achieved CR or PR. | 2.8 [NA to NA] — Ranges for 95% CI were not estimable due to less than 50% participants in this cohort achieved CR or PR. | NA [NA to NA] — Median and ranges for 95% CI were not estimable due to no participants in this cohort achieved CR or PR. | NA [NA to NA] — Median and ranges for 95% CI were not estimable due to no participants in this cohort achieved CR or PR. | NA [NA to NA] — Median and ranges for 95% CI were not estimable due to no participants in this cohort achieved CR or PR.

30. Secondary Outcome: Kaplan-Meier Estimate of Median OS in Part B
Description: OS was defined as time in weeks or months from the start of study treatment to date of death due to any cause. OS was calculated as the death date or last known alive date (if death date unavailable) minus the date of first dose of study medication plus 1 divided by 7 or 30.44 if in months.
Time Frame: Baseline up to 24 months post first dose.
Population: as for outcome 25
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg | Part B2: PF-04518600 30mg + PF-05082566 20mg
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 11 | 30
months | 8.7 [2.4 to 14.3] | 9.5 [3.9 to 22.1] | 12.0 [3.6 to 22.1] | 11.4 [1.3 to 21.1] | 5.4 [1.2 to 11.4] | 12.0 [4.7 to 16.6]

31. Secondary Outcome: Overall Survival Rates at Months 6, 12, and 24 in Part B
Description: Probability of survival at 6, 12, and 24 months after the first dose of study treatment.
Time Frame: Baseline up to 24 months post first dose.
Population: as for outcome 25
Measure: Number (95% Confidence Interval); unit: Probability of survival
Arm/Group | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg | Part B2: PF-04518600 30mg + PF-05082566 20mg
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 11 | 30
Probability of survival
  Survival Probability at Month 6 | 61.4 [26.6 to 83.5] | 61.4 [26.6 to 83.5] | 72.7 [37.1 to 90.3] | 58.4 [22.7 to 82.3] | 45.0 [13.9 to 72.4] | 63.9 [43.2 to 78.8]
  Survival Probability at Month 12 | 30.7 [7.3 to 58.6] | 36.8 [9.3 to 65.7] | 51.9 [19.8 to 76.7] | 43.8 [11.8 to 72.7] | 11.3 [0.6 to 39.1] | 51.9 [31.8 to 68.8]
  Survival Probability at Month 24 | 10.2 [0.6 to 36.4] | 12.3 [0.7 to 41.4] | 20.8 [3.2 to 48.7] | NA [NA to NA] — Number and ranges for 95% CI were not estimable due to all 11 participants in the group have been censored or died before month 24. | 11.3 [0.6 to 39.1] | 6.7 [0.5 to 25.1]

32. Secondary Outcome: Cmax of PF-04518600 Following Single Dose on C1D1 and Css,Max Following Multiple Doses on C3D1 in Part B
Description: as for outcome 14
Time Frame: For Part B1, pre-dose, 1, 4, and 24 hours post dose on C1D1, pre-dose, 1 hour post dose on Day 1 of Cycles 3; For Part B2, pre-dose, 1, and 4 hours post dose on C1D1, pre-dose and 1 hour post dose on Day 1 of Cycles 3.
Population: The PK parameter analysis population was defined as all enrolled participants treated who had sufficient information to estimate at least 1 of the PK parameters of interest. Number of participants analyzed represents the total number of participants in each treatment group in the PK parameter analysis population. Number analyzed represents the number of participants contributing to the summary statistics for Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg | Part B2: PF-04518600 30mg + PF-05082566 20mg
Number analyzed (Participants) | 10 | 12 | 11 | 10 | 9 | 28
µg/mL
  CYCLE1/DAY1 | 2.290 (19) | 6.965 (23) | 7.644 (23) | 19.63 (26) | 62.45 (31) | 10.20 (24)
  CYCLE3/DAY1: number analyzed (Participants) | 9 | 10 | 10 | 8 | 7 | 26
  CYCLE3/DAY1 | 2.779 (29) | 9.049 (21) | 9.359 (31) | 19.76 (45) | 81.49 (51) | 10.53 (39)

33. Secondary Outcome: AUCtau of PF-04518600 Following Single Dose on C1D1 and Following Multiple Doses on C3D1 in Part B
Description: as for outcome 15
Time Frame: as for outcome 32
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg.hr/mL
Arm/Group | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg | Part B2: PF-04518600 30mg + PF-05082566 20mg
Number analyzed (Participants) | 10 | 12 | 11 | 10 | 9 | 28
µg.hr/mL
  CYCLE1/DAY1: number analyzed (Participants) | 9 | 12 | 11 | 10 | 7 | 26
  CYCLE1/DAY1 | 270.7 (27) | 1022 (29) | 1177 (23) | 3089 (19) | 10100 (19) | 1624 (30)
  CYCLE3/DAY1: number analyzed (Participants) | 3 | 7 | 6 | 5 | 5 | 22
  CYCLE3/DAY1 | 340.2 (73) | 1739 (26) | 2239 (18) | 4034 (35) | 19190 (48) | 2291 (45)

34. Secondary Outcome: AUCinf of PF-04518600 Following Single Dose on C1D1 and Following Multiple Doses on C3D1 in Part B
Description: as for outcome 16
Time Frame: as for outcome 32
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*hr/mL
Arm/Group | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg | Part B2: PF-04518600 30mg + PF-05082566 20mg
Number analyzed (Participants) | 10 | 12 | 11 | 10 | 9 | 28
μg*hr/mL
  CYCLE1/DAY1: number analyzed (Participants) | 7 | 2 | 2 | 0 | 1 | 6
  CYCLE1/DAY1 | 283.5 (31) | NA (NA) — Geometric Mean and Geometric CV was not calculated for n<3. And the individual values were 1380,992. | NA (NA) — Geometric Mean and Geometric CV was not calculated for n<3. And the individual values were 1800,1700. |  | 9480 (NA) — Geometric CV was not calculated for n<3. | 1657 (22)
  CYCLE3/DAY1: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0 | 1
  CYCLE3/DAY1 | NA (NA) — Geometric Mean and Geometric CV was not calculated for n<3. And the individual values were 257,228. |  |  | 2710 (NA) — Geometric CV was not calculated for n<3. |  | 1130 (NA) — Geometric CV was not calculated for n<3.

35. Secondary Outcome: t1/2 of PF-04518600 Following Single Dose on C1D1 and Following Multiple Doses on C3D1 in Part B
Description: t1/2 was defined as the time measured for the serum concentration to decrease by one half of the initial concentration.
Time Frame: as for outcome 32
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg | Part B2: PF-04518600 30mg + PF-05082566 20mg
Number analyzed (Participants) | 10 | 12 | 11 | 10 | 9 | 28
days
  CYCLE1/DAY1: number analyzed (Participants) | 7 | 2 | 2 | 0 | 1 | 6
  CYCLE1/DAY1 | 4.104 (1.2263) | NA (NA) — Mean and Standard Deviation was not calculated for n<3. And the individual values were 5.58,5.85. | NA (NA) — Mean and Standard Deviation was not calculated for n<3. And the individual values were 6.98,6.1. |  | 5.61 (NA) — Standard Deviation was not calculated for n<3. | 5.260 (0.76772)
  CYCLE3/DAY1: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0 | 1
  CYCLE3/DAY1 | NA (NA) — Mean and Standard Deviation was not calculated for n<3. And the individual values were 2.72,3.16. |  |  | 4.72 (NA) — Standard Deviation was not calculated for n<3. |  | 3.87 (NA) — Standard Deviation was not calculated for n<3.

36. Secondary Outcome: Cmin of PF-04518600 Following Multiple Doses on C3D1 in Part B
Description: Cmin was defined as Lowest concentration observed during the dosing interval and can be observed directly from data.
Time Frame: as for outcome 32
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg | Part B2: PF-04518600 30mg + PF-05082566 20mg
Number analyzed (Participants) | 9 | 10 | 10 | 8 | 7 | 26
µg/mL | 0.2591 (148) | 2.266 (39) | 1.074 (21520) | 5.327 (101) | 30.59 (38) | 2.671 (155)

37. Secondary Outcome: Cav of PF-04518600 Following Multiple Doses on C3D1 in Part B
Description: Cav was defined as average serum concentration over the dosing interval.
Time Frame: as for outcome 32
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg | Part B2: PF-04518600 30mg + PF-05082566 20mg
Number analyzed (Participants) | 3 | 7 | 6 | 5 | 5 | 22
µg/mL | 1.013 (73) | 5.175 (26) | 6.664 (18) | 12 (35) | 57.15 (48) | 6.815 (45)

38. Secondary Outcome: CL of PF-04518600 Following Multiple Doses on C3D1 in Part B
Description: as for outcome 20
Time Frame: as for outcome 32
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hr/kg
Arm/Group | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg | Part B2: PF-04518600 30mg + PF-05082566 20mg
Number analyzed (Participants) | 3 | 7 | 6 | 5 | 5 | 22
mL/hr/kg | 0.2944 (73) | 0.1725 (26) | 0.1339 (18) | 0.2481 (35) | 0.1566 (48) | 0.1861 (47)

39. Secondary Outcome: Vss of PF-04518600 Following Multiple Doses on C3D1 in Part B
Description: Vss was defined as volume of distribution at steady state.
Time Frame: as for outcome 32
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/kg
Arm/Group | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg | Part B2: PF-04518600 30mg + PF-05082566 20mg
Number analyzed (Participants) | 2 | 0 | 0 | 1 | 0 | 1
mL/kg | NA (NA) — Geometric Mean and Geometric CV was not calculated for n<3. And the individual values were 42.6,46.1. |  |  | 67.4 (NA) — Geometric CV was not calculated for n<3. |  | 54.3 (NA) — Geometric CV was not calculated for n<3.

40. Secondary Outcome: Rac of PF-04518600 Following Multiple Doses on C3D1 in Part B
Description: as for outcome 22
Time Frame: as for outcome 32
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg | Part B2: PF-04518600 30mg + PF-05082566 20mg
Number analyzed (Participants) | 3 | 7 | 6 | 5 | 5 | 22
ratio | 1.374 (31) | 1.593 (26) | 1.762 (12) | 1.361 (37) | 1.861 (31) | 1.413 (31)

41. Secondary Outcome: Cmax of Utomilumab Following Single Dose on C1D1 and Css,Max Following Multiple Doses on C3D1 in Part B
Description: as for outcome 14
Time Frame: as for outcome 32
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg | Part B2: PF-04518600 30mg + PF-05082566 20mg
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 10 | 27
µg/mL
  CYCLE1/DAY1 | 4.018 (33) | 4.06 (39) | 20.33 (43) | 17.63 (33) | 19.02 (29) | 3.232 (22)
  CYCLE3/DAY1: number analyzed (Participants) | 9 | 8 | 11 | 9 | 6 | 26
  CYCLE3/DAY1 | 2.909 (47) | 2.554 (79) | 20.02 (22) | 17.94 (39) | 17.84 (54) | 2.726 (47)

42. Secondary Outcome: AUCtau of Utomilumab Following Single Dose on C1D1 and Following Multiple Doses on C3D1 in Part B
Description: as for outcome 15
Time Frame: as for outcome 32
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg•hr/mL
Arm/Group | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg | Part B2: PF-04518600 30mg + PF-05082566 20mg
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 10 | 27
µg•hr/mL
  CYCLE1/DAY1: number analyzed (Participants) | 10 | 11 | 12 | 9 | 7 | 26
  CYCLE1/DAY1 | 789.4 (23) | 596 (43) | 2465 (33) | 2289 (25) | 2839 (15) | 561.8 (53)
  CYCLE3/DAY1: number analyzed (Participants) | 2 | 4 | 6 | 5 | 4 | 21
  CYCLE3/DAY1 | NA (NA) — Geometric Mean and Geometric CV was not calculated for n<3. And the individual values were 916,464. | 343.7 (225) | 2765 (77) | 673.9 (1191) | 2621 (31) | 232.1 (1524)

43. Secondary Outcome: AUCinf of Utomilumab Following Single Dose on C1D1 and Following Multiple Doses on C3D1 in Part B
Description: as for outcome 16
Time Frame: as for outcome 32
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*hr/mL
Arm/Group | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg | Part B2: PF-04518600 30mg + PF-05082566 20mg
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 10 | 27
μg*hr/mL
  CYCLE1/DAY1: number analyzed (Participants) | 3 | 1 | 9 | 4 | 5 | 5
  CYCLE1/DAY1 | 1011 (20) | 831 (NA) — Geometric CV was not calculated for n<3. | 2801 (25) | 2252 (34) | 3137 (15) | 626.4 (47)
  CYCLE3/DAY1: number analyzed (Participants) | 1 | 0 | 0 | 1 | 2 | 2
  CYCLE3/DAY1 | 467 (NA) — Geometric CV was not calculated for n<3. |  |  | 1950 (NA) — Geometric CV was not calculated for n<3. | NA (NA) — Geometric Mean and Geometric CV was not calculated for n<3. And the individual values were 2360,2970. | NA (NA) — Geometric Mean and Geometric CV was not calculated for n<3. And the individual values were 624,725.

44. Secondary Outcome: t1/2 of Utomilumab Following Single Dose on C1D1 and Following Multiple Doses on C3D1 in Part B
Description: t1/2 was defined as the time measured for the serum concentration to decrease by one half of the initial concentration.
Time Frame: as for outcome 32
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg | Part B2: PF-04518600 30mg + PF-05082566 20mg
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 10 | 27
days
  CYCLE1/DAY1: number analyzed (Participants) | 3 | 1 | 9 | 4 | 5 | 5
  CYCLE1/DAY1 | 11.37 (0.58595) | 5.44 (NA) — Standard Deviation was not calculated for n<3. | 7.769 (2.2299) | 6.873 (1.9954) | 8.27 (2.2945) | 6.632 (2.5566)
  CYCLE3/DAY1: number analyzed (Participants) | 1 | 0 | 0 | 1 | 2 | 2
  CYCLE3/DAY1 | 5.25 (NA) — Standard Deviation was not calculated for n<3. |  |  | 2.59 (NA) — Standard Deviation was not calculated for n<3. | NA (NA) — Mean and Standard Deviation was not calculated for n<3. And the individual values were 13,3.88. | NA (NA) — Mean and Standard Deviation was not calculated for n<3. And the individual values were 5.76,5.8.

45. Secondary Outcome: Cmin of Utomilumab Following Multiple Doses on C3D1 in Part B
Description: Cmin was defined as Lowest concentration observed during the dosing interval and can be observed directly from data.
Time Frame: as for outcome 32
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg | Part B2: PF-04518600 30mg + PF-05082566 20mg
Number analyzed (Participants) | 9 | 8 | 11 | 9 | 7 | 26
µg/mL | 0.03294 (1302300) | 0.002776 (3859511) | 0.08612 (1346874) | 0.0413 (2825205) | 0.3123 (56629) | 0.0007531 (117304)

46. Secondary Outcome: Cav of Utomilumab Following Multiple Doses on C3D1 in Part B
Description: Cav was defined as average serum concentration over the dosing interval.
Time Frame: as for outcome 32
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg | Part B2: PF-04518600 30mg + PF-05082566 20mg
Number analyzed (Participants) | 2 | 4 | 6 | 5 | 4 | 21
µg/mL | NA (NA) — Geometric Mean and Geometric CV was not calculated for n<3. And the individual values were 1.36,0.691. | 0.5119 (225) | 4.119 (77) | 1.004 (1189) | 3.903 (31) | 0.3453 (1524)

47. Secondary Outcome: CL of Utomilumab Following Multiple Doses on C3D1 in Part B
Description: as for outcome 20
Time Frame: as for outcome 32
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hr/kg
Arm/Group | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg | Part B2: PF-04518600 30mg + PF-05082566 20mg
Number analyzed (Participants) | 2 | 4 | 6 | 5 | 4 | 21
mL/hr/kg | NA (NA) — Geometric Mean and Geometric CV was not calculated for n<3. And the individual values were 0.0218,0.04. | 0.05817 (225) | 0.03615 (77) | 0.1483 (1187) | 0.03813 (31) | 0.08619 (1525)

48. Secondary Outcome: Vss of Utomilumab Following Multiple Doses on C3D1 in Part B
Description: Vss was defined as volume of distribution at steady state.
Time Frame: as for outcome 32
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/kg
Arm/Group | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg | Part B2: PF-04518600 30mg + PF-05082566 20mg
Number analyzed (Participants) | 1 | 0 | 0 | 1 | 2 | 2
mL/kg | 6.7 (NA) — Geometric CV was not calculated for n<3. |  |  | 4.22 (NA) — Geometric CV was not calculated for n<3. | NA (NA) — Geometric Mean and Geometric CV was not calculated for n<3. And the individual values were 13.4,4.18. | NA (NA) — Geometric Mean and Geometric CV was not calculated for n<3. And the individual values were 6.46,5.02.

49. Secondary Outcome: Rac of Utomilumab Following Multiple Doses on C3D1 in Part B
Description: as for outcome 22
Time Frame: as for outcome 32
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg | Part B2: PF-04518600 30mg + PF-05082566 20mg
Number analyzed (Participants) | 2 | 4 | 6 | 5 | 4 | 21
ratio | NA (NA) — Geometric Mean and Geometric CV was not calculated for n<3. And the individual values were 1.23,0.493. | 0.5441 (120) | 1.091 (69) | 0.2673 (1381) | 0.9041 (26) | 0.391 (886)

50. Secondary Outcome: Number of Participants With ADA and NAb Against PF-04518600 in Part B
Description: as for outcome 23
Time Frame: Baseline up to end of treatment (maximum of 14 weeks).
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg | Part B2: PF-04518600 30mg + PF-05082566 20mg
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 11 | 30
Participants
  ADA ever-positive: number analyzed (Participants) | 11 | 12 | 12 | 11 | 11 | 28
  ADA ever-positive | 6 | 5 | 3 | 1 | 0 | 13
  NAb ever-positive: number analyzed (Participants) | 11 | 12 | 12 | 11 | 11 | 28
  NAb ever-positive | 1 | 0 | 1 | 0 | 0 | 0

51. Secondary Outcome: Number of Participants With ADA and NAb Against Utomilumab in Part B
Description: as for outcome 23
Time Frame: Baseline up to end of treatment (maximum of 14 weeks).
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg | Part B2: PF-04518600 30mg + PF-05082566 20mg
Number analyzed (Participants) | 10 | 12 | 12 | 9 | 9 | 28
Participants
  ADA ever-positive | 5 | 9 | 9 | 5 | 4 | 22
  NAb ever-positive | 4 | 6 | 7 | 4 | 3 | 22

ADVERSE EVENTS:
Time Frame: AEs: The informed consent date to either 60 days after the last dosing date or the date when all drug-related toxicities are resolved, whichever is later (maximum of approximately 2.25 years for patients in Part A and 3.8 years for patients in Part B). SAEs: The informed consent date to either 98 days after the first dosing date or up to 60 days after the last dosing date, whichever is later (maximum of approximately 2.25 years for patients in Part A and 3.8 years for patients in Part B).
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Part A1: PF-04518600 0.01mg/kg | Part A1: PF-04518600 0.1mg/kg | Part A1: PF-04518600 0.3mg/kg | Part A1: PF-04518600 1.5mg/kg | Part A1: PF-04518600 3.0mg/kg | Part A1: PF-04518600 10mg/kg | Part A2: PF-04518600 30mg | Part A2: PF-04518600 250mg | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg | Part B2: PF-04518600 30mg + PF-05082566 20mg
All-Cause Mortality (participants affected / at risk) | 2/2 | 7/10 | 6/11 | 11/12 | 10/13 | 3/4 | 9/16 | 9/19 | 10/11 | 8/12 | 10/12 | 7/11 | 8/11 | 22/30
Serious Adverse Events (participants affected / at risk) | 0/2 | 4/10 | 1/11 | 3/12 | 6/13 | 2/4 | 7/16 | 6/19 | 5/11 | 2/12 | 3/12 | 5/11 | 5/11 | 10/30
Other Adverse Events (participants affected / at risk) | 2/2 | 10/10 | 11/11 | 12/12 | 13/13 | 4/4 | 16/16 | 19/19 | 11/11 | 12/12 | 12/12 | 11/11 | 11/11 | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A1: PF-04518600 0.01mg/kg (N=2) | Part A1: PF-04518600 0.1mg/kg (N=10) | Part A1: PF-04518600 0.3mg/kg (N=11) | Part A1: PF-04518600 1.5mg/kg (N=12) | Part A1: PF-04518600 3.0mg/kg (N=13) | Part A1: PF-04518600 10mg/kg (N=4) | Part A2: PF-04518600 30mg (N=16) | Part A2: PF-04518600 250mg (N=19) | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg (N=11) | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg (N=12) | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg (N=12) | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg (N=11) | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg (N=11) | Part B2: PF-04518600 30mg + PF-05082566 20mg (N=30)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hernia pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Performance status decreased (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Biliary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Euthanasia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic haemorrhage (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 0.05% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Part A1: PF-04518600 0.01mg/kg (N=2) | Part A1: PF-04518600 0.1mg/kg (N=10) | Part A1: PF-04518600 0.3mg/kg (N=11) | Part A1: PF-04518600 1.5mg/kg (N=12) | Part A1: PF-04518600 3.0mg/kg (N=13) | Part A1: PF-04518600 10mg/kg (N=4) | Part A2: PF-04518600 30mg (N=16) | Part A2: PF-04518600 250mg (N=19) | Part B1: PF-04518600 0.1mg/kg + PF-05082566 20mg (N=11) | Part B1: PF-04518600 0.3mg/kg + PF-05082566 20mg (N=12) | Part B1: PF-04518600 0.3mg/kg + PF-05082566 100mg (N=12) | Part B1: PF-04518600 1.0mg/kg + PF-05082566 100mg (N=11) | Part B1: PF-04518600 3.0mg/kg + PF-05082566 100mg (N=11) | Part B2: PF-04518600 30mg + PF-05082566 20mg (N=30)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 3 | 3 | 1 | 3 | 3 | 0 | 2 | 4 | 3 | 6 | 7
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Deposit eye (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 1 | 3 | 1 | 1 | 3 | 3 | 2 | 1 | 3 | 0 | 1 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 1 | 0 | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 4 | 1 | 3 | 0 | 4 | 0 | 4 | 2 | 2 | 4 | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2 | 4 | 0 | 1 | 1 | 5 | 2 | 1 | 2 | 2 | 1 | 8
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 4 | 1 | 5 | 2 | 1 | 2 | 3 | 4 | 1 | 3 | 1 | 3 | 7
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2 | 2 | 3 | 1 | 2 | 3 | 1 | 1 | 1 | 0 | 3 | 5
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 2 | 0
Catheter site erythema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 2 | 3 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 7 | 6 | 3 | 5 | 1 | 4 | 4 | 1 | 3 | 2 | 3 | 5 | 11
Feeling cold (General disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1
Mass (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1
Oedema (General disorders) | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 2 | 0 | 3 | 0 | 0 | 1 | 3 | 0 | 1 | 1 | 1 | 1 | 3
Pain (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 3 | 2 | 1 | 2 | 1 | 1 | 3 | 0 | 1 | 3 | 3 | 3 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cryptosporidiosis infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 2
Vaginal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 1 | 1 | 1 | 0 | 3 | 2 | 0 | 1 | 1 | 2 | 1 | 5
Amylase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 5 | 1 | 0 | 2 | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 2 | 2 | 1 | 1 | 6 | 7 | 0 | 0 | 1 | 2 | 3 | 4
Basophil count increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 2 | 2 | 1 | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 2
Blood bilirubin increased (Investigations) | 1 | 1 | 0 | 1 | 2 | 0 | 2 | 3 | 0 | 0 | 1 | 0 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 2 | 0 | 2 | 1
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Blood magnesium decreased (Investigations) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram U-wave abnormality (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 4
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 4 | 1 | 1 | 2 | 0 | 0 | 4
Lymphocyte count decreased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Platelet count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Transaminases increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urobilinogen urine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 2 | 1 | 3
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 4 | 1 | 3 | 1 | 5 | 3 | 3 | 3 | 2 | 3 | 4 | 8
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 3
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 3 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 3 | 1 | 2 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 3 | 1 | 0 | 1 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2 | 2 | 0 | 2 | 2 | 2 | 0 | 1 | 0 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 3
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 0
Central nervous system lesion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 2 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 3
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 4 | 1 | 2 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 2
Nervous system disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vasogenic cerebral oedema (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 2 | 3 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 3 | 2
Panic attack (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine flow decreased (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Prostatism (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 2 | 2 | 1 | 1 | 3 | 1 | 2 | 0 | 2 | 2 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 3 | 3 | 1 | 2 | 3 | 2 | 0 | 0 | 2 | 1 | 7
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0/18 | 0 | 0 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Macule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3 | 3 | 3 | 3 | 1 | 2 | 2 | 1 | 1 | 0 | 0 | 1 | 7
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 5 | 3 | 0 | 1 | 2 | 1 | 0 | 3
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 4 | 0 | 0 | 0 | 1 | 1 | 4
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin adhesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperaemia (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 2 | 2 | 1 | 3 | 2 | 0 | 1 | 1 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Intermittent claudication (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Xerophthalmia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1
Medical device site inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatobiliary disease (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asymptomatic bacteriuria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0/1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stoma site discomfort (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Device breakage (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bladder irritation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Embolism venous (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Peripheral coldness (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
A decision was made by the sponsor to terminate further enrollment to the study on 03 Oct 2018 due to business reasons. The decision to terminate study enrollment was not based on any safety or regulatory concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-05-02): https://cdn.clinicaltrials.gov/large-docs/66/NCT02315066/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-12): https://cdn.clinicaltrials.gov/large-docs/66/NCT02315066/SAP_001.pdf